### **Clinical Study Protocol**

| Title | Nabilone for non-motor symptoms in Parkinson's disease: An open-label study to |
|---|---|
| | evaluate long-term safety and efficacy |
| Short Title | The NMS-Nab2 Study |
| Protocol Version | 1.3 |
| Effective | June 2019 |
| Phase | III |
| EudraCT No. | 2017-004253-16 |
| Original Date of Issue | October 2017 |
| Investigational Medicinal Product: | Nabilone: |
| | Synthetic cannabinoid nabilone, other |
| | components: Polyvinylpyrollidone (Povidone) |
| | co-precipitate and corn starch |
| Route and Dosage Form | nabilone 0.25 - 1 mg administered orally once |
| | or twice daily |

#### Confidential Material

The information provided in this clinical investigation plan are strictly confidential and will be available for potential investigators, involved investigators and their study team only, as well as for the medical director of the conducting hospital, health authorities and ethics committees to review, verify or implement the clinical trial. Any publication or disclosure to a third party without prior written consent of the Sponsor is expressly prohibited. By signing the clinical investigation plan, the provisions of it are binding for all parties.

### **General Information**

| Sponsor of the Clinical Trial | Medical University of Innsbruck |
|---|---|
| | Represented by: |
| | O.UnivProf. Dr. Werner Poewe |
| Coordinating Investigator of the Clinical | Department of Neurology Anichstraße 35 6020 Innsbruck Austria E-Mail: mui-sponsor@i-med.ac.at Tel.: 0043-512-504-23850 Fax: 0043-512-504-23852 Prof. Dr. Seppi Klaus |
| Trial | Medical University Innsbruck |
| | Department of Neurology Anichstraße 35 6020 Innsbruck |
| | Austria E-Mail: Klaus.Seppi@tirol-kliniken.at Tel.: 0043-512-504-81498 Fax: 0043-512-504-25819 |
| Author of the Clinical Investigation Plan | Dr. Marina Peball |
| | Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria E-Mail: Marina.Peball@i-med.ac.at Tel.: 0043-512-504-82718 Fax: 0043-512-504-25819 |
| Manufacturer of study medication | AOP Orphan Pharmaceuticals AG |
| | Wilhelminenstraße 91/II<br>1160 Wien<br>Austria<br>Tel.: 0043-1-503 72 44-37 |
| Responsible Contact Person for Drug | Prof. Dr. Hans-Guenther Knaus |
| Safety | Medical University Innsbruck Department for Medical Genetics, Molecular and Clinical Pharmacology Peter-Mayr Strasse 1 A-6020 Innsbruck, Austria Tel.: 0043-512-9003 70440 / 70441 Fax: +43-512-9003 73440 E-mail: hans.g.knaus@i-med.ac.at |

Statistics will be performed by the Study Team.

# Clinical Study Signature Page (1/2)

Title:

Nabilone for non-motor symptoms in Parkinson's disease: An

open-label study to evaluate long-term safety and efficacy

**Short Title:** 

The NMS Nab2 Study

EudraCT-No.:

2017-004253-16

Investigational Medicinal

Product:

Nabilone:

Synthetic cannabinoid nabilone, other components: Povidone

pregelatinized starch, yellow iron oxide (E 172) titanium

dioxide (E 171), gelatin

### Declaration of the Sponsor

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With the signature below the person confirms to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the person agrees to conduct the study as set in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs, if provided and as far as agreed. It has been understood that all documentation previously not published will be kept confidential. Furthermore the person agrees to take all necessary measures to ensure safety and confidentiality of the patient's identities.

O.Univ.-Prof. Dr. Werner Poewe Medical University of Innsbruck Head of the Department of Neurology

Place, Date Signature

# Clinical Study Signature Page (2/2)

# Declaration of the Coordinating Principal Investigator and the Author

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With their signature below the persons confirm to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the persons agree to conduct the study as set put in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs (as far as agreed and provided). It has been understood that all documentation previously not published will be kept confidential. Furthermore the persons agree to keep patient's identities in strictest confidence and to take all required measures to ensure this confidentiality. It is agreed that the Clinical Trial will be conducted according to AMG as well as to the ICH-GCP Guideline (ICH-E6, CPMP/ICH/135/95) and the latest version of the Declaration of Helsinki. To ensure data quality, clinical trial's integrity and compliance with the Clinical Investigation Plan as well as with the various legal and regulatory requirements the Sponsor will visit the participating sites.

With their signature below the person agrees to support visits of authorized persons (e.g. representatives of the Sponsor) and to provide them direct entry to source and other relevant documents in regard to the clinical trial (e.g. CRF, patient files).

Prof. Dr. Seppi Klaus

Medical University of Innsbruck

Principal Investigator

Place, Date, Signature

E PCI

11x 3,11.201

Dr. Marina Peball

Medical University of Innsbruck

Author of the Study Protocol

Place, Date, Signature

# Clinical Study Signature Page, Amendment (1/2)

Title:

Nabilone for non-motor symptoms in Parkinson's disease: An

open-label study to evaluate long-term safety and efficacy

**Short Title:** 

The NMS-Nab2 Study

EudraCT-No.:

2017-004253-16

Investigational Medicinal

Product:

Nabilone:

Synthetic cannabinoid nabilone, other components: Povidone pregelatinized starch, yellow iron oxide (E 172) titanium

dioxide (E 171), gelatin

### Declaration of the Sponsor

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With the signature below the person confirms to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the person agrees to conduct the study as set in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs, if provided and as far as agreed. It has been understood that all documentation previously not published will be kept confidential. Furthermore the person agrees to take all necessary measures to ensure safety and confidentiality of the patient's identities.

O.Univ.-Prof. Dr. Werner Poewe Medical University of Innsbruck Head of the Department of Neurology

Place, Date Signature

# Clinical Study Signature Page, Amendment (2/2)

# Declaration of the Coordinating Principal Investigator and the Author

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With their signature below the persons confirm to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the persons agree to conduct the study as set put in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs (as far as agreed and provided). It has been understood that all documentation previously not published will be kept confidential. Furthermore the persons agree to keep patient's identities in strictest confidence and to take all required measures to ensure this confidentiality. It is agreed that the Clinical Trial will be conducted according to AMG as well as to the ICH-GCP Guideline (ICH-E6, CPMP/ICH/135/95) and the latest version of the Declaration of Helsinki. To ensure data quality, clinical trial's integrity and compliance with the Clinical Investigation Plan as well as with the various legal and regulatory requirements the Sponsor will visit the participating sites.

With their signature below the person agrees to support visits of authorized persons (e.g. representatives of the Sponsor) and to provide them direct entry to source and other relevant documents in regard to the clinical trial (e.g. CRF, patient files).

Prof. Dr. Seppi Klaus Medical University of Innsbruck Principal Investigator

Place, Date, Signature

Dr. Marina Peball

Medical University of Innsbruck

Author of the Study Protocol

1711/2010 A 13.06.202

Place, Date, Signature

# Clinical Study Signature Page, Amendement (1/2)

Title:

Nabilone for non-motor symptoms in Parkinson's disease: An

open-label study to evaluate long-term safety and efficacy

**Short Title:** 

The NMS Nab2 Study

**EudraCT-No.:** 

2017-004253-16

**Investigational Medicinal** 

**Product:** 

Nabilone:

Synthetic cannabinoid nabilone, other components: Povidone

pregelatinized starch, yellow iron oxide (E 172) titanium

dioxide (E 171), gelatin

#### **Declaration of the Sponsor**

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With the signature below the person confirms to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the person agrees to conduct the study as set in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs, if provided and as far as agreed. It has been understood that all documentation previously not published will be kept confidential. Furthermore the person agrees to take all necessary measures to ensure safety and confidentiality of the patient's identities.

O.Univ.-Prof. Dr. Werner Poewe Medical University of Innsbruck Head of the Department of Neurology

Place, Date Signature

# Clinical Study Signature Page, Amendment (2/2)

### Declaration of the Coordinating Principal Investigator and the Author

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With their signature below the persons confirm to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the persons agree to conduct the study as set put in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs (as far as agreed and provided). It has been understood that all documentation previously not published will be kept confidential. Furthermore the persons agree to keep patient's identities in strictest confidence and to take all required measures to ensure this confidentiality. It is agreed that the Clinical Trial will be conducted according to AMG as well as to the ICH-GCP Guideline (ICH-E6, CPMP/ICH/135/95) and the latest version of the Declaration of Helsinki. To ensure data quality, clinical trial's integrity and compliance with the Clinical Investigation Plan as well as with the various legal and regulatory requirements the Sponsor will visit the participating sites.

With their signature below the person agrees to support visits of authorized persons (e.g. representatives of the Sponsor) and to provide them direct entry to source and other relevant documents in regard to the clinical trial (e.g. CRF, patient files).

Prof. Dr. Seppi Klaus

Medical University of Innsbruck

Principal Investigator

Place, Date, Signature

10K 28.11.18

Dr. Marina Peball

Medical University of Innsbruck

Author of the Study Protocol

INNSBRUCK 28-NOV-2

Place, Date, Signature

### Clinical Study Signature Page, Amendment (1/2)

Title: Nabilone for non-motor symptoms in Parkinson's disease: An

open-label study to evaluate long-term safety and efficacy

Short Title: The NMS-Nab2 Study

**EudraCT-No.:** 2017-004253-16

**Investigational Medicinal** 

Product:

Nabilone:

Synthetic cannabinoid nabilone, other components:

polyvinylpyrollidone (Povidone) co-precipitate and corn starch

#### **Declaration of the Sponsor**

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With the signature below the person confirms to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the person agrees to conduct the study as set in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs, if provided and as far as agreed. It has been understood that all documentation previously not published will be kept confidential. Furthermore the person agrees to take all necessary measures to ensure safety and confidentiality of the patient's identities.

O.Univ.-Prof. Dr. Werner Poewe Medical University of Innsbruck Head of the Department of Neurology

Place, Date Signature

### Clinical Study Signature Page, Amendment (2/2)

### Declaration of the Coordinating Principal Investigator and the Author

The present Clinical Investigation Plan was subject to critical review. Its content is consistent with the current risk/benefit evaluation of the IMP as well as with moral, ethical and scientific principles of Good Clinical Practice, the latest version of the Declaration of Helsinki, the local laws and regulations as well as applicable regulatory requirements.

With their signature below the persons confirm to have read this Clinical Investigation Plan and to agree that it contains all information required for study performance. Furthermore, the persons agree to conduct the study as set put in this Clinical Investigation Plan and to adhere to the Sponsor's SOPs (as far as agreed and provided). It has been understood that all documentation previously not published will be kept confidential. Furthermore the persons agree to keep patient's identities in strictest confidence and to take all required measures to ensure this confidentiality. It is agreed that the Clinical Trial will be conducted according to AMG as well as to the ICH-GCP Guideline (ICH-E6, CPMP/ICH/135/95) and the latest version of the Declaration of Helsinki. To ensure data quality, clinical trial's integrity and compliance with the Clinical Investigation Plan as well as with the various legal and regulatory requirements the Sponsor will visit the participating sites.

With their signature below the person agrees to support visits of authorized persons (e.g. representatives of the Sponsor) and to provide them direct entry to source and other relevant documents in regard to the clinical trial (e.g. CRF, patient files).

Prof. Dr. Seppi Klaus

Medical University of Innsbruck

Principal Investigator

Place, Date, Signature

Dr. Marina Peball

Medical University of Innsbruck

Author of the Study Protocol

Place, Date, Signature

134,04-June-loss

# **Study Site and Members of the Study Team**

| Study Site | Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria |
|---|---|
| Members of the Study Team | Prof. Dr. Werner Poewe Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria |
| | Prof. Dr. Klaus Seppi<br>Medical University Innsbruck<br>Department of Neurology<br>Anichstraße 35<br>6020 Innsbruck<br>Austria |
| | Dr. Atbin Djamshidian-Tehrani<br>Medical University Innsbruck<br>Department of Neurology<br>Anichstraße 35<br>6020 Innsbruck<br>Austria |
| | Dr. Marina Peball Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria |
| | Dr. Mario Werkmann<br>Medical University Innsbruck<br>Department of Neurology<br>Anichstraße 35<br>6020 Innsbruck<br>Austria |
| | Dr. Beatrice Heim Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria |
| | Dr. Roberto De Marzi |

Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Philipp Ellmerer Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Federico Carbone Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Kathrin Marini Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Sabine Spielberger Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Olliver Schorr Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dr. Marina Casazza Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Anja Weber, PhD. Medical University Innsbruck

Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Dora Valent, M.Sc. Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

Katarzyna Wachowicz, PhD. Medical University Innsbruck Department of Neurology Anichstraße 35 6020 Innsbruck Austria

### **Additional involved Persons and Institutions**

| | Neurological Study Centre |
|----------------|---------------------------------------------|
| | Medical University of Innsbruck |
| Datamanagement | Anichstraße 35<br>6020 Innsbruck<br>Austria |
| and | |
| Monitoring | Contactperson: |
| Monitoring | Members of the Study team |
| | Tel.: 0043-512 504 - 25810 |
| | Fax: 0043-512 504 - 25819 |
| | E-Mail: |

# **Protocol Synopse**

| Protocol Number: | Version 1.3 |
|---|---|
| Eudract Number: | 2017-004253-16 |
| Study Title: | Nabilone for non-motor symptoms in Parkinson's disease: An open-label study to evaluate long-term safety and efficacy |
| Number of Centers: | One clinical site (Medical University of Innsbruck) |
| Clinical Phase: | III |
| Treatment Duration: | Planned start: April 2018 |
| | Time of Recruitment: 2 months |
| | Titration phase: 2-28 days, 6 months of open-label phase, dose |
| | tapering (individual) and Safety follow-up two weeks after |
| | discontinuation from study drug |
| | Minimum: 186 days / 26 weeks + 4 days |
| | Maximum: 263 days / 37 weeks + 4 days |
| | Planned end of the trial: 2020 (LPLV) |
| Study Population / | Subjects with Parkinson's disease (PD) |
| Indication: | |
| Study Objective: | To test the long-term safety and efficacy of nabilone on non-motor |
| | symptoms (NMS) in subjects with PD |
| Study Design: | Open-label extension study for participants of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial, the NMS-Nab Study. The Safety Follow-Up Visit of the NMS-Nab Study will be the Screening / Baseline Visit of this open-label extension study. Patients will be re-tapered in an open-label nabilone dose optimization phase lasting up to 28 days followed by an open-label period of 6 months on a stable nabilone dose. |
| | the first visit, will be re-tapered with open-label nabilone starting with a dosage of 0.25 mg at the evening. During dose titration and optimization, nabilone will be titrated in 0.25 mg increments (increase by 0.25 mg/ every one to four days), optimally up to the dose the patient had in the open-label titration phase prior to the |

randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial. It is the investigator's decision to modify this dose, if necessary. The retapering will be performed up to a maximum dose of 1 mg twice daily (dose increments: 1: 0.25 mg 0-0-1; 2:

0.25 mg 1-0-1; 3: 0.25 mg 1-0-2; 4: 0.25 mg 2-0-2; 5: 0.25 mg 2-0-3; 6: 0.25 mg 3-0-3; 7: 0.25 mg 3-0-4; 8: 0.25 mg 4-0-4). During titration phase regular two-daily phone calls with the study center will be performed. This open-label titration phase will last up to 28 days and will end with a visit on-site (V 1).

Dose optimization will be assessed with the CGI-I and doses will be adjusted upward in 0.25 mg one to four-daily increments until the patient

- has reached a rating of "1" (i.e. very much improved) or "2" (i.e. much improved) on the 7-point Clinical Global Impression of Improvement (CGI-I; i.e. a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline with the following ratings: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse) [i.e. criterion 1]; or
- experiences intolerable side effects believed to be related to study medication [i.e. criterion 2]; or
- reaches the maximum permitted dosage of 1 mg twice daily [i.e. criterion 3].

#### Patients who meet

- criterion 1 will enter into the 6 months OL treatment period at that dose.
- criterion 2 will proceed to the 6 months OL treatment period at the previous lower dose, providing they will meet the definition of a responder at that dose.
- criterion 3 and were a responder will enter the study at 1 mg twice daily.

Patients are discontinued after dose optimization phase

- if they meet criterion 2 but did not meet the responder definition at the previous dose,
- if they meet criterion 2 at the initial dose of 0.25 mg once daily,
- or if they meet criterion 3 but did not meet the definition of a responder.

Responders will enter the open-label treatment period for 6

months with visits being performed every 3 months in the context of the patient's regularly scheduled visits in the specialized outpatient department. The last visit will be the Termination Visit. Following this, nabilone will be tapered in all patients in 0.25 mg two-daily decrements. During this period the patients will receive phone calls every other day. A Safety Telephone Call and a Safety Follow-Up Visit will be executed 5 days  $\pm$  2 days and 2 weeks  $\pm$  2 days after the last intake of study drug.

#### **Assessments:**

Subjects will be evaluated at the clinic site by the investigator at the Screening / Baseline Visit (ideally Safety Follow-Up of NMS-Nab study), V 1 (end of optimization phase, start of open label nabilone at a fixed dose ranging between 0.25 mg once daily up to 1 mg twice daily), and every 3 months afterwards for 6 months. A Safety Phone Call and a Safety Follow-Up Visit will be performed 5 days  $\pm$  2 days and 2 weeks + 2 days after the end of the last intake of nabilone, respectively.

Study visits will include the following assessments:

- Movement Disorder Society (MDS)-sponsored new version of the UPDRS (MDS-UPDRS) (all visits)
- Non-Motor Symptoms Scale (NMSS) (all visits except for Safety Follow-Up Visit)
- Hospital Anxiety and Depression Scale (HADS) (all visits except for Safety Follow-Up Visit)
- 8-Item Parkinson's Disease Questionnaire (PDQ-8) (all visits except for Safety Follow-Up Visit)
- Montreal Cognitive Assessment Scale (MoCA) (termination visit)
- Mini Mental State Exam (MMSE) (termination visit)
- Epworth Sleepiness Scale (ESS) (all visits except for Safety Follow-Up Visit)
- King's Parkinson's disease pain scale (KPPS) (all visits except for Safety Follow-Up Visit)
- Fatigue Severity Scale (FSS) (all visits except for Safety Follow-Up Visit)
- Columbia Suicide Severity Rating scale (C-SSRS) (all visits)
- CGI-I (V 1, V 2, V 3, and Safety Follow-Up Visit only)
- Vital signs (all visits)
- Concomitant medications (all visits)
- Adverse Events (all visits)
- Physical examination (all visits)
- Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease–Rating Scale (QUIP-RS) (all visits except for Safety Follow-Up Visit)
- Measurement of Eye-Movements with a Tobii TX300 Eye-Tracker (V 2 only)

Subjects will undergo two-daily phone visits during the titration phase and the tapering phase. These will include the following:

- Concomitant medications use
- Adverse Events
- CGI-I
- Hallucination item (1.2) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Day-time sleepiness item (1.8) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Columbia Suicide Severity Rating scale (C-SSRS)

#### **Concomitant medications:**

Anti-parkinsonian treatment:

All anti-parkinsonian medications will be permitted during the study. However, no changes to medications or dosage will be allowed during this trial.

#### Number of subjects:

Maximally 48 responders of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal Study

# Inclusion/ Exclusion criteria:

Subjects must meet all inclusion criteria in order to be eligible for the study:

#### Inclusion criteria:

- In order to be eligible for the study, patients must have completed the double-blind phase of the NMS-Nab trial as responders within the last 2 months.
- For patients that completed NMS-Nab Study over 2 months prior to the Screening Visit, and meet all other inclusion criteria, eligibility should be discussed on a case-by-case basis.
- Only patients without a drug-related SAE or moderate or severe AE during the NMS-Nab Study can be included in the study
- 4. Patients must be able and willing to provide written informed consent prior to any study related procedure

- being performed. Patients with a legal guardian should be consented according to local requirements.
- 5. Patients must be willing and able to take oral medication and able to comply with the study specific procedures.
- 6. The patient is in good health as determined by medical examination.

The inclusion criteria of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial were as follows:

- 1. age ≥30 years
- 2. diagnosis of PD (de novo or on stable medication without disturbing motor fluctuations or dyskinesia)
- NMS with a score of ≥4 on MDS-UPDRS Part 1. One of the following domains have to be affected with a score ≥2: 1.4 (anxious mood) or 1.9 (pain)
- 4. On a stable regimen of anti-parkinson medications for at least 30 days prior to screening and willing to continue the same doses and regimens during study participation
- 5. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation
- 6. Signed a current IRB-approved informed consent form
- 7. Acceptable method of contraception

Any of the following conditions will exclude the subject from entering the study:

 Patients that experienced a drug-related SAE or had a moderate or severe AE during the NMS-Nab Study will be excluded in the study.

The exclusion criteria of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial were as follows:

- 1. Previous participation in any study with nabilone
- 2. current use of cannabinoids or use within 30 days prior to screening
- current or recent (within 30 days prior to screening) participation in another study with an investigational medicinal product
- 4. atypical or secondary parkinsonism

5. presence of motor complications if, based on the investigator's judgment, not adequately controlled (i.e. a score ≥2 on one of the items of the MDS-UPDRS Part IV at screening) 6. Hoehn and Yahr stage ON > 3 7. Evidence of disturbing impulse control disorder 8. History of neurosurgical intervention for PD 9. Presence of clinically significant symptomatic orthostatic hypotension at screening (MDS-UPDRS 1.12 > 210. Use of prohibited medication listed in 7.4.2 11. Laboratory values clinically significant out-of-range at screening or within 4 weeks prior to screening 12. Known or diagnosed sinus tachycardia in ECG evaluation at screening or within 4 weeks prior to screening 13. presence of an acute or chronic major psychiatric disorder (e.g., Major Depressive Disorder, psychosis) or symptom (e.g., hallucinations, agitation, paranoia) (MDS-UPDRS 1.2 and/or 1.3 > 2) 14. recent suicidal attempt within the past five years or suicidal ideation within the past 6 months 15. presence of dementia (MDS-UPDRS 1.1 > 2, MMSE of < 24 at screening) 16. clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation (based on the investigator's judgment). 17. moderate or severe hepatic or renal impairment. 18. History of chronic alcohol or drug abuse within the last 2 years 19. women of child-bearing potential who do not practice an acceptable method of birth control [\*Acceptable methods of birth control for women and men in this study are: surgical sterilization (e.g. tubal ligation for females), intrauterine devices that release hormones (hormone spiral), oral hormonal contraceptive. contraceptive patch, dermal hormonal contraception, vaginal hormonal contraception (NuvaRing®), implants that release progesterone (Implanon®), long-acting injectable contraceptive, partner's vasectomy, a double-protection method, postmenopausal (> 2 year absence of vaginal bleeding).] 20. Pregnant women, or women planning to become pregnant during the course of the study, or nursing women. 21. Known hypersensitivity to any components of the IMP or excipients 22. Patient is legally incapacitated or persons held in an institution by legal or official order 23. Persons with any kind of dependency on the investigator or employed by the Sponsor or investigator Route and Dosage nabilone 0.25 – 1 mg, administered orally once or twice daily Form: **Objectives** The **primary objective** of this study is to evaluate long-term

#### and Endpoints

safety and tolerability of nabilone in PD patients.

The **secondary objectives** of the study are to assess the effects of long-term, open-label dosing with nabilone on different symptoms of PD and quality of life in patients with PD.

#### **Primary Safety and tolerability endpoints:**

- Safety and tolerability will be evaluated with reference to the following:Number of subjects (%) who discontinue the study
- Number of subjects (%) who discontinue the study due to AE
- Adverse Events (AE)
- Physical and neurological examination findings
- Vital signs assessments
- Subjects compliance, prior and concomitant medication use
- Hallucination item (1.2) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Day-time sleepiness item (1.8) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS)

#### **Secondary Efficacy endpoints:**

Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes from V 1 to the termination visit (V 3) in the following assessments:

- Total and different parts of MDS-UPDRS
- Different domains of MDS-UPDRS Part I
- NMSS
- HAD-S
- PDQ-8
- ESS
- FSS
- KPPS
- QUIP-RS
- CGI-I

The change of MMSE and MoCA score values between the Screening Visit of the NMS-Nab Study (before the first intake of nabilone medication) and the termination visit of this study will be assessed as secondary efficacy endpoints.

#### **Exploratory endpoints:**

 Change in reaction time, attention span, and concentrativeness as measured by the Eyetracking examination

#### **Statistical**

#### **Considerations:**

#### Sample size calculation

This is an open-label study. The sample size for this study is not based on statistical considerations; Up to 48 subjects who completed the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and met patient exclusion/inclusion criteria will be enrolled.

#### **Endpoints**

The primary safety analysis will be performed with the safety data set including all patients with the intake of at least one study drug and performing at least V 1. A safety analysis will be performed on all events and tolerability issues, as well as the hallucination item, orthostatic hypotension item, the day-time sleepiness item of Part I of MDS-UPDRS, and C-SSRS occurring through the overall course of the study. This will be a descriptive analysis reporting overall number, frequencies, and percentage of AEs, SAEs, and SUSARs in all patients taking nabilone, patients withdrawn from the study, and patients withdrawn due to an AE. Separate summaries of AEs in regard of severity and relationship to the study drug, separate summaries of AEs leading to withdrawal from the study and separate summaries for SAEs will be provided.

Results of the changes of all clinical scales in this trial will be shown in a descriptive way by median and interquartile range (quartile 1, quartile 3). Mean and standard deviation for the descriptive analysis will also be provided. P-values for the change of the results will be given.

The secondary efficacy criterion will be measured as the change of all assessments between V 1 and month 6. Because an interpolation of data will not be performed in case of a drop-out, the analysis is a per-protocol analysis. All statistical tests will be performed with a two-sided alpha risk of 0.05. For the study's

secondary efficacy analyses, mean changes from V 1 to the 6 months visit will be analyzed by Wilcoxon matched-pairs test. (49) To estimate the treatment effect, we will then compare mean change from V 1 to month 6 visit using analysis of covariance, with value at V 1 as covariate and the treatment group as main effect. Moreover, sensitivity to treatment will be assessed using effect sizes of the different outcome variables when using nabilone to

For CGI-I analyses, distributions of aggregated ratings (amelioration, aggravation) after 6 months will be evaluated by the Wilcoxon matched-pairs test. (49)

treat non-motor symptoms in Parkinson's disease.

For the change in cognition, the score values of MMSE and MoCA will be compared to the values of these scores at the Screening visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study using the Wilcoxon matched-pairs test.

For the Eye-tracking analyses, mean changes from the evaluations of the Screening and the Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study to V 2 of this study will be compared using the Wilcoxon matched-pairs test.

### **List of Abbreviations**

2-AG 2-arachidonoyl glycerol ADR Adverse Drug Reaction

AE An adverse event is "any untoward medical occurrence in a patient or

clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this

treatment". (47)

AMG "Arzneimittelgesetz" = Medicines Act in Austria

Anandamide Arachidonoyl ethanolamide
BID "bis in die" (Latin), twice daily

CA competent authority

cAMP cyclic adenosine monophosphate

CB1 receptor cannabinoid 1 receptor
CB2 receptor cannabinoid 2 receptor

CBD Cannabidiol

CGI-I Clinical Global Impression – Global Improvement

CRF Case Report Form

C-SSRS Columbia Suicide Severity Rating scale

Directive 2001/20/EC Directive 2001/20 der European Commission

DSM-IV Diagnostic and Statistical Manual of Mental Disorders

DSUR Development Safety Update Report

ECG electrocardiogram

ECS endocannabinoid system
ESS Epworth Sleepiness Scale
ET Early Termination Visit

EU European Union

EudraCT European Clinical Trials Database

FAAH fatty acid amide hydrolysis

FSS Fatigue Severity Scale
GCP Good Clinical Practice

GPR55 GTP-binding protein-coupled receptor 55
HADS Hospital Anxiety and Depression Scale

HEENT examination Examination of the head, eyes, ears, nose, throat

HIV Human immunodeficiency virus

ICF Informed Consent Form

ICH International Conference on Harmonisation

IEC/IRB Independent ethics committee/ Institutional review board

IMP Investigational medicinal product

IND Investigational New Drug
ISF Investigator Site File

KPPS King's Parkinson's disease pain scale

LD/CD Treatment Levodopa / Carbidopa Treatment

LID Levodopa-induced Dyskinesia

LPLV Last Patient Last Visit

MDS Movement Disorder Society

mg Milligramme mm Millimetre

MMSE Mini Mental State Examination

MoCA Montreal Cognitive Assessment Scale

MS Motor symptoms

NMS Non-motor symptoms

NMSS Non-Motor Symptoms Scale

OFF state the phase with no response to medication and significant motor symptoms

OH orthostatic hypotension

OL open-label

ON state period when the patient notices a benefit on MS from standard oral LD/CD

treatment

PD Parkinson's disease

PDQ-8 8-Item Parkinson's Disease Questionnaire
PPAR peroxisome proliferator-activated receptor

QUIP-RS Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease—

Rating Scale

RBD REM Sleep Behavior Disorder
RCT randomized controlled trials

REM rapid eye movement

RNA Ribonucleic acid

SAE "A serious adverse event (experience) or reaction is any untoward medical

occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in

persistent or significant disability/incapacity, or is a congenital

anomaly/birth defect". (47)

SOP Standard Operating Procedures

SUSARs A SUSAR is an event that is believed to be causal to the to the

administration of the study drug and is severe and unexpected.

TMF Trial Master File
TC Telephone Call

TC – S Safety Telephone Call

TRPV1 transient receptor potential vanilloid type 1 cation channel

UPDRS Unified Parkinson Disease Rating Scale

V Visit

V – S Safety Follow-Up Visit

VAS of Pain Visual Analog Scale of Pain

 $\Delta^9$ -THC  $\Delta^9$  – tetrahydrocannabinol

#### **Table of contents**

| G | eneral | Information | 2 |
|---|---|---|---|
| CI | inical | Study Signature Page (1/2)Fehler! Textmarke nicht | definiert. |
| CI | inical | Study Signature Page (2/2)Fehler! Textmarke nicht | definiert. |
| St | udy S | ite and Members of the Study Team | 6 |
| Αc | ditio | nal involved Persons and Institutions | 14 |
| | | I Synopse | |
| | | Abbreviations | |
| 1 | | kground and Rationale | |
| | 1.1 | The endocannabinoid system | |
| | 1.2 | Non-motor symptoms in Parkinson's Disease | |
| | 1.3 | Preclinical Research in Parkinson's disease | 35 |
| | 1.4 | Therapeutic potential of Cannabinoids in Parkinson's Disease | 35 |
| 2 | Obj | ectives and Endpoints | 37 |
| | 2.1 | Objectives | 37 |
| | 2.1. | 1 Primary Objectives | 37 |
| | 2.1. | 2 Secondary Efficacy Objectives | 37 |
| | 2.1. | 3 Exploratory Objective | 38 |
| | 2.2 | Endpoints | 38 |
| | 2.2. | 1 Primary Endpoints | 38 |
| | 2.2. | 2 Secondary Efficacy Endpoints | 38 |
| | 2.2. | 3 Exploratory Endpoints | 38 |
| 3 | Stu | dy Design | 39 |
| | 3.1 | Study Description | 39 |
| | 3.1. | 1 Study end: | 40 |
| | 3.1. | 2 Visits | 41 |
| | 3.1. | Study Duration Per Patient | 42 |
| | 3.1. | Planned Number of Patients | 42 |
| | 3.1. | 5 Anticipated Regions and Countries | 43 |
| | 3.2 | Schedule of Events | 44 |
| | 3.3 | Schematic Diagram | 45 |
| 4 | Stu | dy Population and Withdrawal of Patients | 46 |
| | 4.1 | Inclusion Criteria | |

| | 4.2 | Exclusion Criteria | 47 |
|---|---|---|---|
| | 4.3 | Discontinuation of the Study, Premature Termination | 48 |
| | 4.3 | .1 Potential Criteria for Withdrawal from Study | 49 |
| | 4.3 | .2 Definite Criteria for Withdrawal from Study | 49 |
| | 4.4 | Further treatment after end of treatment | 50 |
| | 4.5 | Closure of the Study | 50 |
| 5 | Stu | ıdy Procedures (by Visits) | 51 |
| | 5.1 | Recruitment and Screening / Baseline Visit | 51 |
| | 5.1 | .1 Recruitment and Informed Consent Process | 51 |
| | 5.1 | .2 Screening / Baseline Visit (V 0) | 53 |
| | 5.2 | Dose Titration Phase | 54 |
| | 5.3 | Visit V 1 | 55 |
| | 5.4 | Visit V 2 | 5 <i>6</i> |
| | 5.5 | Termination Visit / V 3 | 57 |
| | 5.6 | Safety Telephone Call (TC – S) and Safety Follow-Up Visit (V – S) | 59 |
| | 5.7 | Early Termination Visit | |
| | 5.8 | Unscheduled Visit / USV | 60 |
| | 5.9 | Telephone calls | 61 |
| 6 | De | scription of Assessments: Efficacy and Safety Variables | 62 |
| | 6.1 | Secondary Endpoints: Assessments of Efficacy | |
| | 6.2 | Primary Endpoints: Safety Assessments | 66 |
| | 6.2 | .1 Adverse Events, Serious Adverse Events, Adverse Drug Reaction, Suspected | |
| | une | expected serious adverse reactions | 66 |
| | 6.2 | .2 Description of other safety measures | 67 |
| | 6.3 | Assessment of exploratory endpoint | 68 |
| 7 | Stu | ıdy Treatments | 70 |
| | 7.1 | Details of Study Treatment | |
| | 7.1 | | |
| | | 70 | |
| | 7.1 | | 70 |
| | 7.1 | <u> </u> | |
| | 7.1 | | |
| | 7.2 | Subject's Compliance | |
| | 7.2 | | |
| | 7.3 | Drug Accountability and Treatment Compliance | |
| | 73 | 1 Procedures for Monitoring Patient Compliance | 72 |

| | <b>7.4</b> | Prior and Concomitant Medications/Treatments | 73 |
|---|---|---|---|
| | 7.4. | 1 Allowed Anti-PD Medications/Treatments | 73 |
| | 7.4. | Prohibited Concomitant Medications/Treatments | 73 |
| | 7.5 | Concomitant Non-Pharmacologic Therapies | 74 |
| 8 | Adv | /erse Events | 75 |
| | 8.1 | Summary of known and possible Adverse Events of the IMP | 75 |
| | 8.2 | Definition of an Adverse Event (AE) | 76 |
| | 8.3 | Definition of a Serious Adverse Events (SAEs) | 77 |
| | 8.4 | Adverse Drug Reaction (ADR) & Unexpected Adverse Drug Reaction | 78 |
| | 8.5 | Suspected Unexpected Serious Adverse Reactions (SUSARs) | 79 |
| | 8.6 | Pregnancy | 79 |
| | 8.7 | Overdose of Investigational Medicinal Product | 80 |
| | 8.8 | Grading of Severity of Adverse Events | 80 |
| | 8.9 | Causality | 81 |
| | 8.10 | Recording, Reporting, and Follow-Up Procedures | 82 |
| | 8.10 | Procedures for Recording, Reporting, and Follow-Ups of Adverse Events | 82 |
| | 8.10 | | |
| | Sus | pected Unexpected Serious Adverse Reactions | 83 |
| | 8.11 | Review and Annual report on Adverse Events, Serious Adverse Events and | |
| | Suspe | cted Unexpected Serious Adverse Reactions | 85 |
| 9 | Do | cumentation | 87 |
| | 9.1 | Data Recording (Case Report Form, CRF and Patient's Record) | 88 |
| | 9.2 | Trial Folders | 89 |
| | 9.2. | 1 Trial Master File (TMF) | 89 |
| | 9.2. | 2 Investigator Site File (ISF) | 90 |
| | 9.3 | Data Storage | |
| | 9.3. | | |
| | 9.3. | 2 Storage duties of the investigator | 90 |
| 1 | 0 E | ata Management | 91 |
| 1 | 1 P | rotocol Deviations | 91 |
| 1: | 2 S | tatistical Analysis | 92 |
| | 12.1 | Determination of Sample Size | |
| | 12.2 | Study Populations: Datasets or Populations analyzed | |
| | 12.3 | Background and Demographic Characteristics | |
| | 12.4 | Safety Analysis | |
| | 12.5 | Efficacy Variables and Analysis | 94 |

| 12.6 | Exploratory Endpoint | 94 |
|------|------------------------------------------------------|-----|
| 12.7 | Handling of Missing Data | 94 |
| 13 | Quality Management | 96 |
| 13.1 | Qualifications | 96 |
| 13.2 | Monitoring | 96 |
| 13.3 | Audits and Inspections | 97 |
| 14 | Reporting | 98 |
| 14.1 | Annual Progress Reports | 98 |
| 14.2 | Final Study Report | 98 |
| 15 | Publication | 99 |
| 16 | Amendments | 99 |
| 17 | Ethical and Regulatory Aspects | 100 |
| 17.1 | Responsibilities of the Sponsor and the investigator | 100 |
| 17.2 | Approval and Consent | 101 |
| 17.3 | Patient Insurance | 103 |
| 17.4 | Data Protection and Confidentiality | 103 |
| 17.5 | Discontinuation of the Study by the Sponsor | 104 |
| 18 | References | 105 |
| 19 | Index of Figures | 109 |
| 20 | Index of Tables | 109 |

### 1 Background and Rationale

### 1.1 The endocannabinoid system

The endocannabinoid system (ECS) has become a center of attention for its (neuro)modulatory effects in the last 25 years and has become a potential target of drug therapy for a variety of illnesses. The ECS plays an important role in many physiological body functions and influences mood, motor control, cognition, eating behavior, and nociception. Therefore, indications like neuropathic pain, anorexia, and spasticity associated with multiple sclerosis or spinal trauma, as well as chemotherapy-induced emesis can now be treated with cannabinoids like nabilone, dronabinol, sativex, and epidiolex. [12,31,32]

The two main cannabis species *sativa* and *indica* have been the ancestors of almost all strains that exist today and from which more than 60 pharmacologically active components derive. The main psychoactive compound of *Cannabis sativa* is  $\Delta^9$  – tetrahydrocannabinol ( $\Delta^9$ -THC), which has a stronger euphoric potential than isolated components of Cannabis indica that have more sedative, analgesic, and antiemetic effects. [1,12]

The ECS summarizes endogenous cannabinoids (endocannabinoids), cannabinoid receptors and their synthesis, and degradation enzymes.

Endocannabinoids are endogenous lipids and ligands to cannabinoid receptors. Arachidonoyl ethanolamide (anandamide) and 2-arachidonoyl glycerol (2-AG) have been the first discovered and therefore best known endogenous cannabinoids out of a large group of molecules binding to the endocannabinoid receptors. Endocannabinoids are not stored in vesicles like other neurotransmittors. They show a release on-demand into the extracellular space mainly through retrograde signaling after postsynaptic activation with the duty to decrease presynaptic neurotransmission. After their local and short-lasting task is fulfilled endocannabinoids are taken up by surrounding cells and degraded mainly by fatty acid amide hydrolysis (FAAH) for anandamide and by monoacylglycerol lipase for 2-AG. [2,12,32]

The endocannabinoid receptors, named CB1 and CB2, are G-protein coupled, seven-transmembrane domain receptors of the Gi and Go classes. Both are activated mainly by cannabinoids and their synthetic analogues, eicosanoids or aminoalkylindoles as well as by a large number of synthesized agonists, inverse agonists, antagonists and allosteric modulators. [1] Activation of these receptors inhibits adenylate cyclases and subsequently increases the intracellular amount of cyclic adenosine monophosphate (cAMP), resulting in alteration of the level of activity in voltage- dependent calcium channels and potassium channels and an activation of several mitogen-activated protein kinases. [3]

The CB1 cannabinoid receptor is referred to as the "brain cannabinoid receptor" due to its numerous occurrence in all brain structures. Particularly, the Cortex, Basal Ganglia, Hippocampus and Cerebellum present with a high density of CB1 receptor. Combining all its effects, the CB1 receptor aids in the control of cell survival, differentiation and proliferation, and several cell functions. Through retrograde activation the duration of synaptic activation, synaptic plasticity, and neurotransmitter release is influenced. [1,4,32]

Moreover, non-neuronal cells of the brain, astrocytes in particular, express the CB1 receptor in a large amount and its activation through glutamate release leads to an activation of presynaptic metabotropic glutamate receptor. [5]

The occurrence of the CB1 receptor is not limited to the brain, but also appears in the peripheral nervous system and other mammal tissues and organs, where it aids in maintaining homeostasis. [1]

The CB2 receptor is of little homology to the CB1 receptor but shows similar ways of activation through Gi/o. It is expressed mostly in cells and organs playing a role in the body's immune system where its activation reduces the liberation of pro-inflammatory response (cytokines, lymphoangiogenic factors). [6] CB2 receptors are also expressed in the gastrointestinal tract and in microglia and vascular cells of the brain as well as in the dorsal vagal motor nucleus, the nucleus ambiguous and the spinal trigeminal nucleus. CB2 receptor activation may contribute to affective behavior but its concrete role in the brain is not defined yet. In the gastrointestinal tract effects on food intake, gastrointestinal motility, gastric secretion and gastroprotection, cell proliferation, and intestinal inflammatory processes are discussed. [7]

In 2003 the U.S. Health and Human Services granted U.S. Patent 6630507 which describes the use of components extracted from Cannabis sativa as useful in neuroprotective disorders like PD, Alzheimer's disease, and HIV- induced dementia. [33] Neuroprotective potential of cannabinoids is believed to be due to receptor- induced but also – independent mechanisms and specific effects of several endocannabinoids and synthetic agents, like THC, CBD, cannabinol, CP55,940, and AM404 (an anandamide analog). [12] In preclinical experiments, cannabinoids have the ability to counteract reactive oxygen species and strengthen endogenous antioxidants and thereby prevent oxidative stress on neuronal cells by reducing microglial and proinflammatory activation through agonistic action of the CB2 receptor system as well as by reducing glutamatergic excitotoxicity. [34, 12]

Moreover, there exist other receptors where several endocannabinoids like anandamide can bind to under certain circumstances, like the transient receptor potential vanilloid type 1 (TRPV1) cation channel, the peroxisome proliferator-activated receptor (PPAR), the

abnormal-CBD receptor and the GTP-binding protein-coupled receptor (GPR)55 that possibly influence the clinic of movement disorders. [1,12]

**Nabilone** is an analogue of dronabinol (THC), the psychoactive component of cannabis, but it is not derived from the cannabis plant in contrast to dronabinol. Nabilone acts as a partial agonist on both CB1 and CB2 receptor in humans and therefore mimics the effect of THC but with more predictable side effects and less euphoria. In Austria, nabilone is licensed for the use as an antiemetic for chemotherapy-induced nausea and vomiting not responding to conventional antiemetic treatment. The FDA approved nabilone for treating anorexia and weight loss in patients with AIDS. Nabilone is widely used as an adjunct therapy for chronic pain management, although it is only officially approved for this use in Mexico. Nabilone is a racemate consisting of the (S,S) and the (R,R) isomers ("trans") with an average weight of 372.5408 Dalton. After oral administration it is rapidly absorbed via the gastrointestinal tract. The major excretory pathway is the biliary system. The half-life of nabilone amounts to 2 hours, with a half-life of its metabolites of around 35 hours. The chemical formula of nabilone is:  $C_{24}H_{36}O_3$ .

### 1.2 Non-motor symptoms in Parkinson's Disease

Parkinson's Disease (PD) is a neurodegenerative disorder that occurs with a prevalence of 1,6/1000 in both males and females equally in all geographical areas. It is less common in Asia than in Europe, Africa, North America, South America, or Australia and its prevalence is increasing with age (1% in 60 years old people, 3% at the age of 80 years). The mean age of onset is 55 years (17 – 80 years).

Although PD is generally considered a paradigmatic movement disorder, it has long been recognized that the neuropathology underlying PD involves many brain areas that are not directly involved in motor control. [14,15] It is therefore not surprising that a majority, if not all, PD patients suffer from non-motor symptoms adding to the overall burden of parkinsonian morbidity. [16,17,18] In this trial, male and female PD patients without disturbing motor fluctuations or dyskinesia over the age of 30 years suffering from non-motor symptoms (measured on the basis of UPDRS Part I, including at least anxiety or pain) will be included. Non-motor symptoms in PD involve a multitude of functions including disorders of sleep-wake cycle regulation, cognitive dysfunction, disorders of mood and affect, autonomic dysfunction as well as sensory symptoms and pain. They become increasingly prevalent and obvious over the course of the illness and are a major determinant of quality of life, progression of overall disability, and of nursing home placement in PD. [19]

Common non-motor symptoms in late stage PD include hallucinations, dementia, and

autonomic dysfunction including urinary incontinence, constipation, and symptomatic

orthostatic hypotension. In PD patients who have had 20 years of disease duration, dementia occurs in 83%, hallucinosis in 74%, symptomatic OH in 48%, constipation requiring daily laxatives in 40% and urinary incontinence in 71%. [18]

Moreover, certain non-motor symptoms such as constipation, olfactory loss, anxiety, depression, and RBD may antedate the onset of classical motor symptoms by years or even decades. [20,21,22,23,24,25,26]

Unlike most motor features of PD, NMS often have limited treatment options or response. [13] Although common, there is a paucity of research concerning the diagnosis and treatment of non-motor symptoms in PD. Indeed, non-motor symptoms in PD are frequently missed or undeclared during routine consultations and well-performed large-scale RCTs for the treatment of the different non-motor symptoms in PD are lacking. [27,28]

However, a variety of treatments are available, and for some patients, these treatments can effectively control or improve disability from non-motor symptoms, such as psychiatric symptoms, sleep disorders, autonomic dysfunction, and fatigue (see Table 1).

Table 1: Drug classes for non-motor symptoms in PD

| NON-MOTOR SYMPTOMS | DRUG CLASS (NAME) |
|---|---|
| Disorders of sleep and wakefulness | |
| REM Sleep behavioural disorder | Benzodiazepine (Clonazepam), hormons (Melatonin) |
| Autonomic dysfunction | |
| Constipation | Osmotic laxative (Polyethylene Glycol),<br>Chloride channel activator (Lubiprostone) |
| Gastrointestinal motility | Peripheral dopamine antagonist (Domperidone) |
| Orthostatic hypotension | Peripheral dopamine antagonist (Domperidone), mineralcorticoid (Fludrocortisone), vasopressor (Midodrine), acetylcholineesterase inhibitor (Pyridostigmine), Norepinephrine prodrug (Droxidopa) |
| Sialorrhoea | Anticholinergic (Atropine drops,<br>Glycopyrrolate), Neurotoxin (Botulinum toxin<br>A, Botulinum toxin B) |
| Cognitive impairment | |
| Dementia | Acetylcholinesterase inhibitor (Rivastigmine) |
| Psychiatric symptoms | |
| Depression | Dopamine agonist (Pramipexole), serotonin reuptake inhibitor / serotonin and norepinephrine reuptake inhibitor (Citalopram, Escitalopram, Fluoxetine, Paroxetine, Sertraline, Venlafaxine extended release), Tricyclic antidepressant (Desipramine, Nortriptyline) |
| Psychosis | Atypical antipsychotic (Clozapine, Quetiapine), Acetylcholinesterase inhibitor (Rivastigmine) |
| Other | Fatigue (Stimulant Methylphenidate, Modafinil) |

#### 1.3 Preclinical Research in Parkinson's disease

The endocannabinoid system (ECS) functions as a regulator of dopamine release and uptake. Inversely, changes of dopamine levels in the brain can alter the ECS. [9,10] To date the hypothesis is that endocannabinoids are a compensational mechanism to the loss of dopamine in patients with PD. [1,12] A reduction of CB1 receptors has been shown in post mortem analyses of the caudate nucleus, anterior dorsal putamen and external segment of the globus pallidus in comparison to normal levels to the rest of the brain. This might be related to an overactive endocannabinoid system with increased CB1 receptor activity, messenger RNA levels and levels of endocannabinoids in the basal ganglia which has been described in animal models. It is believed that these findings play a role in motor symptoms of patients with PD and can be influenced by Levodopa therapy. [1,11,30] Moreover, neuroprotective properties of cannabinoids in preclinical experiments are gaining more and more attention for clinicians dealing with patients with movement disorders. These effects are mainly due to antioxidant mechanisms, microglial inhibition and modulation of cell-cell interaction of glia cells and neuronal cells in the basal ganglia. [1,11,30]

Indeed, activated microglia have been found in lesions of neurodegeneration in the substantia nigra of deceased patients with PD in comparison to healthy person. Moreover, a decrease of microglial activation is the reason why CB2 receptor agonists have shown to reduce inflammation and degeneration of dopaminergic neurons in PD. [1,11,30] Interestingly, Barrero et. al discovered that polymorphisms in the cannabinoid receptor gene influence depressive mood in patients with PD. [35]

# 1.4 Therapeutic potential of Cannabinoids in Parkinson's Disease

The endocannabinoid system takes part in building emotions, motor control, attention and concentration, the sensation of pain, and eating. [12,31,32]

Evidence of effects of cannabinoids on symptoms in PD from clinical trials is scarce. Most of these trials are either small-sized with less than 20 patients included [12,40,42] or uncontrolled [12,36,37,38,39].

Improvement of motor and non-motor symptoms in PD after intake of cannabinoids has been described in several uncontrolled observational studies with ameliorated rest tremor, bradykinesia, rigidity, and Levodopa-induced Dyskinesia (LID) as well as improved pain, psychosis, symptoms of RBD, and sleep-quality. These effects could not be reproduced by randomized controlled trial (RCTs), which were small-sized and used different cannabinoids.

Thus, while a randomized, double-blind, placebo-controlled crossover trial in 7 PD patients suggested improvement of Levodopa-induced Dyskinesia (LID) with the synthetic cannabinoid nabilone (0.03mg/kg nabilone per day) [42], another randomized, double-blind, placebo-controlled crossover trial in 19 PD patients found no effects on LID with an oral cannabis extract (40). Interestingly the same study did not show any effects on QoL (40), while another parallel-group randomized controlled trial (RCT) [43] in 21 PD patients treated with placebo, cannabidiol (CBD) 75 mg/day or CBD 300 mg/day reported improved QoL in patients using CBD 300 mg/day and placebo. The same study showed no difference in the mean total UPDRS scores of patients with placebo and CBD in different dose regimens. Overall, there is no conclusive evidence from RCT on the symptomatic treatment of motor symptoms in PD. [12,40, 43, 42]

Cannabinoids were well tolerated in all of these trials. No serious adverse events were recorded. The most common side effects from the RCTs have been the feeling of dizziness in up to 10% of patients, mild hypotension in up to 90% of patients, deterioration or new-onset change of perception (hallucinations, the feeling to be detached, confusion), and somnolence in up to 47% of patients. [40,42, 43] In one RCT two patients withdraw from the study due to vertigo and postural hypotension resulting from receiving nabilone but this was not consistent with other RCTs which included a greater sample size and documented no withdrawals due to side effects of cannabinoids.

Due to the overall impact of NMS in PD and based on the influence of the endocannabinoid system on NMS in broad manner in PD, we decided to perform a proof of concept study to test nabilione for the treatment of NMS in PD.

We hypothesize that because of the described effects of the endocannabinoid system, nabilone will improve non-motor symptoms in patients with PD. This therapy should be well tolerated by contrast to some of the drug classes used in standard medical care and can therefore be an ethically justified additional treatment option for symptoms not concerning motor control of PD. If the treatment shows to be effective, the use of nabilone in health care practice can be supported by the data from this study.
#### 2 Objectives and Endpoints

#### 2.1 Objectives

#### 2.1.1 Primary Objectives

The **primary objective** of this study is to evaluate safety and tolerability of nabilone in PD patients.

Safety and tolerability will be evaluated with reference to the following:

#### 1. Tolerability

- Number of subjects (%) who discontinue the study
- Number of subjects (%) who discontinue the study due to AE
- 2. Safety Measures
- Adverse Events (AE)
- Physical and neurological examination findings
- Vital signs assessment including performance of active orthostatism (measurement of heart rate and blood pressure after 10 minutes of quiet rest in the supine position and at 1, 2, 3, 5, and 10 minutes of active standing)
- Subjects compliance
- Prior and concomitant medication use
- Hallucination item (1.2) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society – Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Day-time sleepiness item (1.8) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS)

#### 2.1.2 Secondary Efficacy Objectives

The **secondary objectives** of the study are to assess the effects of long-term, open-label dosing with nabilone concerning non-motor symptoms and quality of life in patients with PD.

Long-term efficacy evaluations are the secondary objective of this study. Efficacy endpoints include changes from V 1 to the termination visit in the following assessments:

- Total and different parts of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Different domains of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I
- Non Motor Symptoms Scale (NMSS)
- Hospital anxiety and depression scale (HAD-S)
- Parkinson's Disease Questionnaire 8 (PDQ-8)
- Epworth Sleepiness Scale (ESS)

- Fatigue Severity Scale (FSS)
- King's Parkinson's disease pain scale (KPPS)
- Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease–Rating Scale (QUIP-RS)
- Clinical Global Impression Global Improvement (CGI-I)

The change of MMSE and MoCA score values between the Screening Visit of the NMS-Nab Study (before the first intake of nabilione medication) and the termination visit of this study will be assessed as secondary efficacy endpoints.

#### 2.1.3 Exploratory Objective

The exploratory objective of this study will be an Eye-tracking evaluation in PD patients taking nabilone at Visit V 2:

 Change of the reaction time, attention span, and concentrativeness between Screening and Termination Visit of the randomized placebocontrolled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and V 2 of this study as measured by the Eye-tracking examination.

#### 2.2 Endpoints

#### 2.2.1 Primary Endpoints

The primary endpoint will be the long-term safety and tolerability of nabilone between V 1 and the termination visit using measures described in 2.1.1.

#### 2.2.2 Secondary Efficacy Endpoints

The change in all other assessments listed above between V 1 and the termination visit will be the secondary efficacy criteria, as well as the MoCa and MMSE as compared to the values at Screening of the NMS-Nab Study.

#### 2.2.3 Exploratory Endpoints

The change of the reaction time, attention span, and concentrativeness between Screening and Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and V 2 of this study as measured by the Eye-tracking examination will be an exploratory endpoint.

#### 3 Study Design

#### 3.1 Study Description

This is a mono-centric Phase III, open-label study in patients with Parkinson's disease formerly participating in the randomized placebo-controlled, double-blind, parallel-group phase of the enriched enrolment randomized withdrawal trial NMS-Nab Study. Optimally, the Safety Follow-Up Visit of the NMS-Nab Study will be the Screening / BaselineVisit of this open-label extension study. Patients will be re-tapered in an open-label nabilone dose optimization phase lasting up to 28 days followed by an open-label period of 6 months on a stable nabilone dose.

Patients must meet all inclusion criteria and none of the exclusion criteria. Eligible subjects, who have signed the informed consent form at the first visit, will be re-tapered with open-label nabilone starting with a dosage of 0.25 mg at the evening. During dose titration and optimization, nabilone will be titrated in 0.25 mg increments (increase by 0.25 mg/ every one to four days), optimally up to the dose the patient had in the open-label titration phase prior the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial. It is the investigator's decision to modify this dose, if necessary. The re-tapering will be performed up to a maximum dose of 1 mg twice daily.

The dose increments will be hold as follows:

```
1. 0.25mg 0-0-1;
```

- 2. 0.25mg 1-0-1;
- 3. 0.25mg 1-0-2;
- 4. 0.25mg 2-0-2;
- 5. 0.25mg 2-0-3;
- 6. 0.25mg 3-0-3;
- 7. 0.25mg 3-0-4;
- 8. 0.25mg 4-0-4.

Regular **phone calls** with the study center will be performed every other day during titration phase. These will include the following:

1. Concomitant medications use, 2. Adverse Events, 3. CGI-I, 4. Hallucination item (1.2), Orthostatic hypotension (OH) item (1.12), Day-time sleepiness item (1.8) of MDS-UPDRS 5. C-SSRS

The open-label titration phase will last up to 28 days and ends with an on-site visit (V 1). Afterwards, patients will be on a stable nabilone dose for 6 months.

Dose adjustments during titration phase will be performed until the patient:

- 1. has much (CGI-I Rating Scale: 2) or very much (CGI-I Rating Scale: 1) improved NMS on the 7-point Clinical Global Impression of Improvement Scale.
- 2. experiences intolerable side effects believed to be related to the study medication or;
- 3. reaches the maximum permitted dosage of 1 mg twice daily.

Criterion 1 defines responders. Patients who meet this criterion will enter into the open-label treatment period at the last prescribed dose. Patients who meet criterion 2 will proceed to the open-label treatment period at the previous lower dose, providing they will meet the definition of a responder at that dose. Patients who meet criterion 3 and were responder will enter the study at 1 mg twice daily.

Patients are discontinued after dose optimization phase if they meet criteria number 2 but did not meet the responder definition at the previous dose, if they meet criteria 2 at the initial dose of 0.25 mg once daily, or if they meet criteria 3 but did not meet the definition of a responder.

During the open-label treatment period, dose adjustments can be performed if CGI-I deteriorates. In this case, patient will re-enter the titration phase of the trial.

After the dose optimization visit, the patient will enter the 6 months open-label treatment period with nabilone in the dose defined in the titration phase. Visits will be performed every 3 months (V 2, V 3) in the scope of the patients regular visits in the specialized outpatient department. V 3 will be the termination visit. Following this, nabilone will be tapered in all patients in 0.25 mg two-daily decrements. Phone calls will be held every other day during dose tapering phase. The patients will be asked for the use of concomitant medications, AEs, CGI-I, the items 1.2, 1.8, and 1.12 of MDS-UPDRS Part I, and the C-SSRS. A phone call for safety issues will be held after 5 days  $\pm$  2 days and a Safety Follow- Up Visit will be scheduled after 2 weeks + 2 days of discontinuation from study drug. (see 5.6)

#### 3.1.1 Study end:

1) After having finished the 6 months of open-label treatment phase, patients will be down-titrated from the study medication in 0.25 mg decrements every other day. During tapering two-daily phone calls will be held, asking for concomitant medications, AEs, CGI-I, the items 1.2, 1.8, and 1.12 of MDS-UPDRS Part I, and the C-SSRS. A safety call will be performed 5 days ± 2 days after having stopped study medication and a safety follow-up visit will be done 2 weeks + 2 days after having stopped study medication. (see 5.6) If there should be deterioration of parkinsonism

- or non-motor features, the patients should be offered prescription of a cannabinoid drug.
- 2) If the trial is stopped on behalf of the Sponsor or a regulatory authority or if patients withdraw from study medication due to personal or medical reasons during the course of the study, the patients will be advised to come to the hospital as soon as possible for an Early Termination Visit (see 5.7). A Safety Follow-Up Visit should be performed 2 weeks + 2 days after the last intake of study medication (if the Early Termination Visit occurs not longer than 5 days after the discontinuation of the study medication). (for reasons for discontinuation and withdrawal see 4.3, for ET and Safety Follow-Up Visit see 5.6)

#### **3.1.2 Visits**

Subjects will be evaluated in the study center by the investigator at the Screening / Baseline Visit, at the end of the open-label titration phase (i.e. V 1), and every 3 months ( $\pm 7$  days) afterwards (V 2 at month 3  $\pm 7$  days, V 3 at month 6  $\pm 7$  days). A Safety Telephone Call (TC – S) and Safety Follow- Up Visit (V - S) will be performed 5 days  $\pm$  2 days and 2 weeks + 2 days after the last intake of study drug.

The following scales or questionnaires will be performed during all study visits:

- Movement Disorder Society (MDS) sponsored new version of the UPDRS (MDS-UPDRS) (all visits)
- 2. Non-Motor Symptoms Scale (NMSS) (all visits except for Safety Follow-Up)
- 3. Hospital Anxiety and Depression Scale (HADS) (all visits except for Safety Follow-Up)
- 4. 8-Item Parkinson's Disease Questionnaire (PDQ-8) (all visits except for Safety Follow-Up)
- 5. Montreal Cognitive Assessment Scale (MoCA) (termination visit)
- 6. Mini Mental State Exam (MMSE) (termination visit)
- 7. Epworth Sleepiness Scale (ESS) (all visits except for Safety Follow-Up)
- 8. King's Parkinson's disease pain scale (KPPS) (all visits except for Safety Follow-Up)
- 9. Fatigue Severity Scale (FSS) (all visits except for Safety Follow-Up)
- 10. Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease–Rating Scale (QUIP-RS) (all visits except for Safety Follow-Up)
- 11. Columbia Suicide Severity Rating scale (C-SSRS) (all visits)
- 12. Clinical Global Impression Global Improvement (V 1, V 2, V 3, and Safety Follow-Up Visit only)
- 13. Vital signs (all visits)
- 14. Concomitant medications (all visits)

- 15. Adverse Events (all visits)
- 16. Physical and neurological examination (all visits)
- 17. Measurement of Eye-Movements with a Tobii TX300 Eye-Tracker (V 2 only)

#### 3.1.3 Study Duration Per Patient

Recruitment will start after the ethical committee and regulatory authorities approve the study and all necessary documents are available and filed. Recruitment phase will last to the point when all of the 48 patients of the double- blind phase of the NMS-Nab trial have been asked if they are willing to participate in this extension trial.

The study will begin with the Screening / Baseline Visit. If a patient is eligible for the study, he/she will then enter the open-label dose titration phase. This optimization phase will last from 2 up to 28 days for each patient and will include phone calls every other day and a visit at the end of the titration phase (V 1). The patients will stay on the open-label medication for 6 months which ends with the termination visit. Afterwards, the nabilone dose will be tapered and a Safety Follow-Up will be performed via telephone call and on-site visit.

The total anticipated study duration for an individual patient starting from the Screening / Baseline Visit will be a minimum of 186 days / 26 weeks + 4 days (including safety follow-up visit) and a maximum of 263 days / 37 weeks + 4 days. The end of the study is defined as the date of the last visit of the last patient in the study (LPLV).

#### 3.1.4 Planned Number of Patients

This is an open-label study. The sample size for this study is not based on statistical considerations; Up to 48 subjects who completed the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and met patient exclusion/inclusion criteria will be enrolled.

In the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study a total of 38 patients provided 80% power at a 2-sided 5% significance level to detect a statistically significant difference in the change from randomization to Week 4 in MDS-UPDRS Part I score between nabilone and placebo if the true difference is 2.5 points. In the absence of previous data, we empirically chose as clinically meaningful a 2.5 units change from randomization to the visit at 4 weeks (in Phase 2). This sample size calculation assumed a standard deviation of the change from randomization to week 4 to be 2.4 points. (46) Assuming a drop-out rate of 25%, we planned to include around 48 patients with Parkinson's disease in the NMS-Nab trial.

Importantly, although a sample size calculation is provided, this was an exploratory study evaluating different NMS domains. Furthermore, corrections for multiple comparisons are therefore not planned.

# 3.1.5 Anticipated Regions and Countries This study will be held at one clinical site (Medical University of Innsbruck).

#### 3.2 Schedule of Events

Table 2: Nabilone for non-motor symptoms in Parkinson's Disease

| STUDY<br>PERIOD | Screening /<br>Baseline | Dose<br>Titrati<br>on<br>Period | Open-label Phase | | | Dose Tapering | | Safety<br>Follow-<br>Up | Early<br>Terminat<br>-<br>ion |
|---|---|---|---|---|---|---|---|---|---|
| STUDY<br>PERIOD | Screening /<br>Baseline | Dose<br>Titratio<br>n<br>Phase | Open-label<br>Phase | | | | | | |
| STUDY<br>WEEK,<br>STUDY<br>VISIT | Week 0,<br>Screening /<br>Baseline<br>Visit | Tele-<br>phone<br>calls | Monat 0, Visite<br>1 | Monat 3,<br>Visite 2 | Monat 6,<br>Visite 3,<br>Termination<br>Visit | Tele-<br>phone<br>calls | Safety<br>Follow-<br>Up Phone<br>Call | Safety<br>Follow-Up<br>Visit<br>V - S | Early<br>Terminat-<br>ion Visit<br>ET |
| Visit<br>Descriptor | V 0 | | V 1 | V 2 | V 3 | | | V - S | ET |
| Visit<br>window<br>(days) | Day 0 | Every<br>other<br>day | month 1 ±<br>7 days | 3 months<br>± 7 days | 3 months<br>± 7 days | Every<br>other day<br>until IMP<br>Stopp | 5 days ±<br>2 days<br>after IMP<br>Stopp | 2 weeks +<br>2 days<br>after IMP<br>Stopp | As soon<br>as<br>possible<br>after the<br>last intake<br>of IMP |
| Written<br>Informed<br>consent | Х | | | | | | | | |
| Vital signs <sup>1</sup> | Х | | Х | Х | Х | | | Х | Х |
| Adverse<br>Events | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Con-<br>comitant<br>Medication | Х | Х | Х | Х | Х | X | Х | Х | Х |
| Physical<br>and Neurol.<br>Exam | Х | | Х | Х | Х | | | Х | Х |
| Urine<br>pregnancy<br>test | Х | | Х | Х | Х | | | | Х |
| MDS-<br>UPDRS | Х | Partly<br>(Part<br>I) | Х | Х | Х | Partly<br>(Part I) | Partly<br>(Part I) | Х | Х |
| NMSS | Х | -/ | Х | Х | Х | | | | Х |
| HADS | Х | | Х | Χ | Х | | | | Х |
| PDQ-8 | Х | | Х | Х | Х | | | | Х |
| MoCA | | | | | Х | | | | Х |
| ESS | X | | X | Χ | Х | | | | Х |
| KPPS | Х | | X | Х | Х | | | | Χ |
| FSS | X | | X | Х | Х | | | | Х |
| CGI-I | | Х | Х | Х | Х | Х | Х | Х | Х |
| MMSE | | | | | Х | | | | Х |
| C-SSRS | X | Х | X | Х | Х | Х | Х | Х | Х |
| QUIP-RS | Х | | Х | Х | Х | | | | Х |
| Eye-<br>tracking | | | | Х | | | | | Х |
| Dispense<br>IMP | Х | | Х | Х | Х | | | | |
| Drug<br>Account-<br>ability | | | X | Х | Х | | | Х | Х |

<sup>&</sup>lt;sup>1</sup> Vital Signs include height (only at Screening / BaselineVisit), weight, temperature, pulse rate and blood pressure after at least 10 minutes of rest and at 1,3,5, and 10 minutes of active standing.

#### 3.3 Schematic Diagram



Figure 1: Schematic Diagram for participants

#### 4 Study Population and Withdrawal of Patients

#### 4.1 Inclusion Criteria

In order to be eligible for participation in the study, subjects must meet all inclusion criteria:

- 1. In order to be eligible for the study, patients must have completed the double-blind phase of the NMS-Nab trial as responders within the last 2 months.
- 2. For patients that completed NMS-Nab Study over 2 months prior to the Screening / Baseline Visit, and meet all other inclusion criteria, eligibility should be discussed on a case-by-case basis.
- Only patients without a drug-related SAE or moderate or severe AE during the NMS-Nab Study can be included in the study
- 4. Patients must be able and willing to provide written informed consent prior to any study related procedure being performed. Patients with a legal guardian should be consented according to local requirements.
- 5. Patients must be willing and able to take oral medication and able to comply with the study specific procedures.
- 6. The patient is in good health as determined by medical examination and based on the investigator's judgement

The inclusion criteria of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial were as follows:

- 1. Age ≥30 years
- 2. Diagnosis of PD: PD should be either de novo or on stable medication without disturbing motor fluctuations or dyskinesia.
- 3. NMS with a score of ≥4 on MDS-UPDRS Part 1. One of the following domains have to be affected with a score ≥2: 1.4 (anxious mood) or 1.9 (pain)
- 4. On a stable regimen of anti-parkinson medications for at least 30 days prior to screening and willing to continue the same doses and regimens during study participation
- 5. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation
- 6. Patient is informed and had enough time and opportunity to think about his/her participation in the study and has signed a current IRB-approved informed consent form
- 7. Contraception
  - a. Women of childbearing potential must use or attest an acceptable method\* of contraception starting 4 weeks prior to study drug administration and for a minimum of 1 month after study completion.
  - b. Men with a potentially fertile partner must be willing to use an acceptable method\* of contraception for the duration of the study and for 3 months after study drug discontinuation or have had a vasectomy.

\*Acceptable methods of birth control for women and men in this study are: surgical sterilization (e.g. tubal ligation for females), intrauterine devices that release hormones (hormone spiral), oral hormonal contraceptive, contraceptive patch, dermal hormonal contraception, vaginal hormonal contraception (NuvaRing®), implants that release progesterone (Implanon®), long-acting injectable contraceptive, partner's vasectomy, a double-protection method, postmenopausal (> 2 year absence of vaginal bleeding). This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus). The regulations for contraception are derived from Guideline ICH E8 Chapter 3.2.2.1 Selection of subjects together with ICH M3 Note 4.

#### 4.2 Exclusion Criteria

Patients with any of the following characteristics will be excluded from entering the study:

- 1. Patients with PD who have not participated in the randomized double-blind phase of the previous NMS-Nab Study.
- 2. Patients that experienced a drug-related SAE or had a moderate or severe AE during the NMS-Nab Study will be excluded in the study.
- 3. Patients who are unable or unwilling to comply with the study procedures in the investigator's opinion.
- 4. Patients with any clinically significant or unstable medical or surgical condition at the Screening / Baseline Visit that may preclude safety and the completion of the study participation (based on the investigator's judgement).

The exclusion criteria of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal trial were as follows:

- 1. Patient previously participated in any study with nabilone.
- 2. Current use of cannabinoids or use of cannabinoids within 30 days prior to screening.
- 3. Patient is currently participating in or has participated in another study of investigational products within 30 days prior to screening.
- 4. Patient has any form of secondary or atypical parkinsonism (e.g., drug-induced, post stroke).
- 5. Patient presents with motor complications which are, based on the investigator's judgment, not adequately controlled (i.e. a score ≥2 on one of the items of the MDS-UPDRS Part IV at screening)
- 6. Hoehn and Yahr stage > 3
- 7. Evidence of disturbing (i.e. requiring treatment) impulse control disorder in the participant. Can be resolved through a structural interview during screening period.
- 8. History of neurosurgical intervention for PD
- presence of symptomatic orthostatic hypotension at screening (MDS-UPDRS 1.12 > 2)
- 10. Use of prohibited medication listed in 7.4.2
- 11. Patients with laboratory values that are out-of-range at Screening (or within 4 weeks prior to Screening) and haven't been reviewed and documented as not clinically significant by the investigator. Lab Tests can be repeated for confirmation.
- 12. Patients with known or newly diagnosed sinus tachycardia in ECG evaluation at Screening or within 4 weeks prior to Screening.

- 13. presence of an acute or chronic major psychiatric disorder (e.g., Major Depressive Disorder, psychosis) or symptom (e.g., hallucinations, agitation, paranoia) (MDS-UPDRS 1.2 and/or 1.3 > 2)
- 14. Patients who had a recent suicidal attempt (active, interrupted, aborted) within the past five years or report suicidal ideation within the past 6 months.
- 15. presence of dementia (MDS-UPDRS 1.1 > 2, MMSE of <24 at the Screening visit)
- 16. Clinically significant or unstable medical or surgical condition at Screening or Baseline visit that may preclude safety and the completion of the study participation (based on the investigator's judgement).
- 17. Patients with moderate or severe hepatic or renal impairment.
- 18. Patient has a history of chronic alcohol or drug abuse within the last 2 years.
- 19. women of child-bearing potential who do not practice an acceptable method of birth control (See: acceptable methods of birth control at 4.1.)
- 20. Pregnant women or women planning to become pregnant during the course of the study and nursing women.
- 21. Patients who are knowingly hypersensitive to any of the components of the IMP or excipients.
- 22. Patient is legally incapacitated or persons held in an institution by legal or official order
- 23. Persons with any kind of dependency on the investigator or employed by the Sponsor or investigator

#### 4.3 Discontinuation of the Study, Premature Termination

Subjects have the right to withdraw fully or partially from the study at any time and for any reason without prejudice to their future medical care by the physician or at the institution. Withdrawal of full consent for a study means that the subject does not wish to receive further investigational treatment and does not wish or is unable to continue further study participation. Subject data up to withdrawal of consent will be included in the subject's study data, but no further information will be collected unless a separate consent has been given. Withdrawal of partial consent means that the subject does not wish to take the protocol-specified product any longer but is still willing to collaborate in providing further data by continuing on study.

**The investigator** has the right to discontinue a patient from IMP or withdraw a patient from the study at any time. The primary reason for withdrawal from the study should be documented. Patients should be discontinued if they experience intolerable side effects believed to be related to the study drug and they will be terminated if they did not meet the responder criterion at the previous dose or the maximum permitted dose.

The **Sponsor** has the right to discontinue this trial at any time. The Sponsor will notify the investigator if the sponsor decides to stop the clinical trial.

The Sponsor has the right to terminate the trial prematurely at any time.

This might be if there are any relevant medical or ethical concerns, or if completing the trial is no longer practicable. If such action is taken, the reasons for terminating the trial must be documented in detail. All trial subjects still under treatment at the time of termination must undergo a final examination (Early Termination Visit as soon as possible and Safety Follow-

Up Visit 2 weeks + 2 days after the ET (if the ET is performed after 5 days after the last intake of study drug)) which must be documented. The principal investigator must be informed without delay if any investigator has ethical concerns about continuation of the trial. In case of discontinuation of the trial the IEC and competent regulatory authority must be informed within 15 days of early termination.

#### 4.3.1 Potential Criteria for Withdrawal from Study

The investigator should inform the Monitor if any of the following events occur that may lead to a discontinuation of the participation in the study:

- 1. Noncompliance of the patient with the study procedures or medications.
- 2. The patient doesn't have a stable PD or changes his/her medication or receives neurosurgical intervention for PD.
- 3. The patient presents with one or more clinically significant laboratory values that are not within normal limits or clinically significant abnormal findings on physical examination, or experiences AEs that are intolerable (as determined by the patient) or that endanger the safety of the patient based on the investigator's judgement.

#### 4.3.2 Definite Criteria for Withdrawal from Study

A definite withdrawal from the study must be operated if any of the following events occur:

- 1. The patient withdraws his/ her consent willingly.
- 2. Patient develops a psychiatric, medical or surgical condition that would interfere with his/ her participation.
- 3. Patient shows abnormal laboratory values concerning hepatic and renal function as described in the exclusion criteria.
- 4. Pregnancy of the patient during the study, as confirmed by a positive pregnancy test.
- 5. Withdrawal of the patient is requested by the Sponsor or a regulatory agency.
- 6. The Sponsor or a regulatory agency discontinues the study. Reasons for discontinuation may include, but are not limited to the following:
  - Patient enrolment is unsatisfactory
  - Administrative Reasons
- 7. The Sponsor terminates the study prematurely. Premature termination of the trial will be considered if:
  - The risk-benefit balance for the trial subject changes markedly.
  - It is no longer ethical to continue treatment with the IMP.
  - The Sponsor considers that the trial must be discontinued for safety reasons.
  - An interim analysis or results of other research show that one of the trial treatments is superior or inferior to another.
  - It is no longer practicable to complete the trial.
- 8. Patient has performed an active suicide since the last visit or reports any suicidal behavior. In this case he/she should be referred to a hospital for Mental Health immediately.

Should the trial be discontinued or should a subject request or decide to withdraw from the study, all efforts will be made to complete and report the observations as thoroughly as possible up to the end of withdrawal.

Thus, if a discontinuation of or a withdrawal from the study occurs, all observations, evaluations as well as lab results and other test results should be documented. Moreover, a

short description of the primary reason(s) for removing the patient must be recorded in the source documents and provided to the Sponsor.

In case of a discontinuation of or a withdrawal from the study every effort should be made for attendance of an Early Termination (ET) Visit, which will be scheduled as soon as possible, followed by a Safety Follow-Up Visit after 2 weeks + 2 days of the ET (if the ET is performed after 5 days after the last intake of study drug) (see 5.6 and 5.7). Patients will not be followed for any reason after consent has been withdrawn, unless a separate consent has been given for further data collection.

In case the withdrawal was due to an AE the patient should be followed up until he/she has recovered/ it has resolved, has reached a stable state, the investigator determines that it is no longer clinically significant, or the patient is lost to follow up. (see 8)

#### 4.4 Further treatment after end of treatment

After the end of the study treatment, alternative methods for the therapy of disturbing non-motor symptoms in PD can be prescribed to the patients as seen in Table 1: Drug classes for non-motor symptoms in PD, keeping in mind the patient's tolerance. If the patient has shown benefit from the therapy with nabilone, a cannabinoid therapy will be prescribed on behalf of the investigator's decision.

#### 4.5 Closure of the Study

The clinical trial shall be deemed to end when the last patient absolved the planned last visit according to protocol. The completion of the study will be reported to the ethics committee as well as to the relevant authorities.

#### 5 Study Procedures (by Visits)

An overview of the study procedures, including the time of events and assessments performed, may be found in 3.2 and 3.3. Details of scales used to evaluate efficacy and safety can be found in Section 6.1 and 6.2 and in the applicable appendices. A detailed description of study procedures by visit will be provided in this section.

Eligible subjects who meet all inclusion criteria and none of the exclusion criteria at the Screening / Baseline Visit will be titrated to the optimal dose as described above which could last up to 28 days. During this phase regular phone calls will be held every other day. After reaching the optimal dose, the patients will visit the outpatient clinic for an on-site visit (V 1) and enter the 6 months of open-label treatment phase with 4-monthly visits. The first dose of IMP will be taken at home after the Visit V 1. A Safety Phone call will take place 5 days ± 2 days and a Safety Follow-Up visit will be performed 2 weeks + 2 days after the last intake of study medication. At visits after intake of medication, the patients will be requested to return the IMP kits (including all used, unused, and partially used medication) dispensed to them at the previous visit and to take their IMP in the morning before every visit. Furthermore, the patients should take their concomitant medication at home and at the clinic, if permitted, as normally scheduled. Safety evaluations will be performed as scheduled in the schedule of events table with examination of vital signs, AE, concomitant medication, the items 1.2, 1.8, and 1.12 of MDS-UPDRS Part I, and the C-SSRS operated at every visit and AE and concomitant medication, the items 1.2, 1.8, and 1.12 of MDS-UPDRS Part I, and the C-SSRS at every phone call. In the event of Early Termination, patients will be asked to complete an Early Termination Visit as soon as possible and to return for a Safety Follow-Up Visit 2 weeks + 2 days after their last dose of IMP.

Please refer to the Schedule of Events table and the Schematic diagram (in 3.2 for specific timing of assessments and Section 5.1,5.2,5.3,5.4,5.5,5.6,5.7, , and 6 for a detailed description of timing and aim of study procedures and scales.

#### 5.1 Recruitment and Screening / Baseline Visit

#### 5.1.1 Recruitment and Informed Consent Process

Patients previously participating in the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal NMS-Nab Study will be seen in the outpatient department on-site or at the neurologic wards.

The Screening / Baseline Visit of this study may coincide with the Safety Follow-Up Visit of the NMS-Nab study. If the Screening / Baseline Visit occurs on the same day as the last visit of the NMS-Nab study, procedures or assessments completed for the NMS-Nab study do not need to be repeated for this trial.

For interested patients a member of the qualified research team will explain the study purpose, goals, and requirements in an understandable way and an IRB/IEC-approved informed consent form will be handed to the patients considering participation for information. Relevant contact from the site including phone numbers will be given to the patient. Thus the patient can read, ask questions, and consult his/her family members if requested. It is the responsibility of the principal investigator, or a subinvestigator delegated by the principal investigator to obtain written informed consent from each subject prior to participation in the trial, following adequate explanation of the aims, methods, anticipated benefits and potential hazards of the study. The person taking consent must be GCP trained, suitably qualified and experienced, and have been delegated this duty by the PI on the delegation log.

The investigator or designee will explain the patients are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason. No clinical trial procedures will be conducted prior to taking consent from the participant. Consent will not denote enrolment into trial.

If all questions are clarified and the patient has been given ample time to think about his/her participation, the informed consent will be obtained in accordance with ICH GCP by signing the informed consent form at a visit on-site before any trial-related procedures are completed. The signature from the investigator who conducted the informed consent discussion and the patient as well as the date will be provided and documented in the source documents. For patients who consent to participate in the study a copy of the signed ICF and other information available will be provided to them prior to participation. The original signed and dated ICF will be maintained at the investigator's site.

Any patient who is unable to demonstrate understanding of the information contained in the ICF won't be allowed to participate in the study. The ICF and any other information provided to patients will be revised whenever important new information (e.g. safety information resulting in significant changes in the risk/benefit assessment) becomes available that is relevant to the consent and continued participation of a patient in the study. The revised ICF and information must receive IRB/IEC-approval prior to its use, and a copy of the IRB/IEC's approval will be provided to the Sponsor. The patient will be informed of any new information via the revised ICF or information material by the investigator and his/her willingness to further participate in the study will be questioned. A signed and dated new ICF will be obtained and stored, and a copy will be given to the patient. This will as well be recorded in the source documents.

After providing and documenting consent on the IRB/IEC-approved written ICF, patients will be enrolled into the NMS-Nab2 study and will continue with their assigned subject identification number from the NMS-Nab study.

#### 5.1.2 Screening / Baseline Visit (V 0)

All subjects must provide written informed consent before any study-specific assessments or procedures are performed.

The following assessments will be performed during the Screening / Baseline Visit and used to determine whether a patient is eligible for the study or not.

If the NMS-Nab2 Screening / Baseline Visit occurs on the same day as the last visit of the NMS-Nab Study, procedures or assessments completed for the NMS-Nab Study do not need to be repeated for this Screening / Baseline Visit.

#### **Screening / Baseline Assessments:**

- 1. Obtain written informed consent (see Section 5.1.1), sign and date, and provide a copy to the patient.
- 2. review inclusion and exclusion criteria for eligibility
- 3. review demographics, medical, medication and psychiatric history, review neurological and PD history, including questions for disturbing (i.e. treatment required) impulse control disorders and anti-PD medications.
  - a. If less than 2 months have passed between the patient's completion of the NMS-Nab Study and the Screening / Baseline Visit, and there are no changes to medical, medication, or psychiatric history since completion of the NMS-Nab study, these data do not have to be re-captured.
  - b. If the gap is more than 2 months, the information has to be re-captured.
- 4. Perform assessment of Vital signs: obtain weight, height, and temperature, obtain and record serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing
- 5. Urine sample for pregnancy test (for women of childbearing potential only)
- 6. Perform brief physical and neurological examination (see: 6.2.2)
- 7. Administer the MDS-UPDRS Part I, II, III, and IV (record if patient is in ON or OFF state), and the Modified Hoehn and Yahr stage.
- 8. Administer the following assessments:
  - a. NMSS
  - b. HADS
  - c. PDQ-8
  - d. ESS

- e. FSS
- f. KPPS
- g. C-SSRS
- h. QUIP-RS

If the patient does not meet eligibility criteria at the time of screening, e.g., if an unstable medical condition disqualifies the patient from participating in the study, the patient is considered a screen failure. Record the primary reason for screen failure in the source documents.

Screen failures maybe eligible for rescreening to acceptable parameters. This will need to be discussed with the Sponsor or designee.

Screening does not necessarily constitute enrolment of the subject.

- 9. Dispense the IMP kits to the patient so that he/she has enough until the –next Visit.
- 10. Record the dates the patient is instructed to take the study drug on the packaging of it. Record the following information in the source documents: patient number, IMP kit number, date, and time the study drug was dispensed.
- 11. Instruct the patient to bring his/her used, unused, and partially used IMP kits to the next visit and schedule this visit.
- 12. Review the dosing instructions for the study drug with the patient and answer any questions. The patient will be instructed to take one tablet of the study drug by mouth two times daily starting in the evening after the Screening / Baseline Visit. The evening dose should be approximately 12 hours after the morning dose. Document that the patient understood the dosing instructions.

#### **5.2 Dose Titration Phase**

For patients who remain eligible, proceed with starting nabilone with a dosage of 0.25 mg in the evening and titrate in in one- to four-daily increments at a maximum dosage of 1 mg twice daily. Optimally, the dose will be increased until the dose the patient was a responder in the NMS-Nab study. It is the investigator's decision to adapt this dose.

Dose increments will be held as follows:

1. 0.25 mg 0-0-1; 2. 0.25 mg 1-0-1; 3. 0.25 mg 1-0-2; 4. 0.25 mg 2-0-2; 5. 0.25 mg 2-0-3; 6. 0.25 mg 3-0-3; 7. 0.25 mg 3-0-4; 8. 0.25 mg 4-0-4.

Regular **phone calls** with the study center will be performed every other day during titration phase. These will include questions for concomitant medication, AEs, and the assessment of

the CGI-I. Moreover, the items 1.2, 1.8, and 1.12 of MDS UPDRS Part I, and the C-SSRS will be assessed. The duration of the open-label titration phase can range from 2 days up to 28 days.

Dose adjustments during titration phase will be performed until the patient:

1. Criterion 1: has much (CGI-I Rating Scale: 2) or very much (CGI-I Rating Scale: 1) improved NMS on the 7-point Clinical Global Impression of Improvement Scale.

This criterion defines responders. Patients who meet this criterion will enter into the 4-weeks treatment period at the last prescribed dose.

2. Criterion 2: experiences intolerable side effects believed to be related to the study medication.

Patients who meet criteria 2 will proceed to the 4-weeks treatment period at the previous lower dose, assuming they will meet the definition of a responder at that dose.

3. Criterion 3: reaches the maximum permitted dosage of 1 mg twice daily.

Patients who meet criteria 3 and were a responder will enter the study at 1 mg twice daily.

Patients are discontinued if they meet criteria number 2 but did not meet the responder definition at the previous dose, if they meet criteria 2 at the initial dose of 0.25 mg once daily, or if they meet criteria 3 but did not meet the definition of a responder.

#### 5.3 Visit V 1

Patients will have an on-site visit at the clinic after they meet the responder criterion at their "optimal dose". The following assessments should be performed at this visit:

- 1. Perform assessment of Vital signs: obtain weight and temperature, obtain and record serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing
- 2. Ask for AE occurring since the last visit.
- 3. Interview on concomitant medication use since the last visit.
- 4. Urine sample for pregnancy test (for women of childbearing potential only)
- 5. Perform physical and neurological examination
- 6. Administer the MDS-UPDRS Part I, II, III, and IV (record if patient is in ON or OFF state), and the Modified Hoehn and Yahr stage
- 7. Administer the following assessments:
  - a. NMSS
  - b. HADS
  - c. PDQ-8
  - d. ESS

- e. FSS
- f. KPPS
- g. CGI-I
- h. C-SSRS
- i. QUIP-RS
- 8. Collect all used, unused, and partially used study drug and record it in the source documents and Drug Accountability Section.
- 9. Schedule the next visit, which must occur after 3 months  $\pm$  7 days on stable nabilone dosage from the date of the Visit 1.
- 10. Instruct the patient to bring their medication to the next visit (including concomitant medication so that they are able to maintain their regular treatment schedule)
- 11. Dispense the IMP kits assigned by the Sponsor to the patient so that he/she has enough until the next Visit.
- 12. Record the dates the patient is instructed to take the study drug on the packaging of it. Record the following information in the source documents: patient number, assigned IMP kit number, date, and time the study drug was dispensed.
- 13. Review the dosing instructions for the study drug with the patient, answer any questions, and remind the patient to return all used, unused, and partially used study drugs at the next visit. The patient will be instructed to take the pre-specified number of tablets of the study drug by mouth two times daily starting in the evening after this Visit. The evening dose should be approximately 12 hours after the morning dose. Document that the patient understood the dosing instructions.

The patient will leave the clinic with enough IMP for the next 3 months  $\pm$  7 days and begin to take the assigned IMP (nabilone) in the evening after this visit.

#### 5.4 Visit V 2

The visit V 2 will be held 3 months  $\pm$  7 days after the Visit V 1. The following assessments should be performed and documented with date and time at this on-site visit:

- 1. Perform assessment of Vital signs: obtain weight, temperature, obtain and record serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing
- 2. Ask for AE occurring since the last visit.
- 3. Interview on concomitant medication use since the last visit.
- 4. Urine sample for pregnancy test (for women of childbearing potential only)
- 5. Perform physical and neurological examination

- 6. Administer the MDS-UPDRS Part I, II, III, and IV (record if patient is in ON or OFF state), and the Modified Hoehn and Yahr stage
- 7. Administer the following assessments:
  - a. NMSS
  - b. HADS
  - c. PDQ-8
  - d. ESS
  - e. FSS
  - f. KPPS
  - g. CGI-I
  - h. C-SSRS
  - i. QUIP-RS
  - j. Eye-tracking
- 8. Collect all used, unused, and partially used study drug and record it in the source documents and Drug Accountability Section.
- 9. Schedule the next visit, which must occur after 3 months  $\pm$  7 days on stable nabilone dosage from the date of the Visit V 2.
- 10. Instruct the patient to bring their medication to the next visit (including concomitant medication so that they are able to maintain their regular treatment schedule)
- 11. Dispense the IMP kits assigned by the Sponsor to the patient so that he/she has enough until the next Visit.
- 12. Record the dates the patient is instructed to take the study drug on the packaging of it. Record the following information in the source documents: patient number, assigned IMP kit number, date, and time the study drug was dispensed.
- 13. Review the dosing instructions for the study drug with the patient, answer any questions, and remind the patient to return all used, unused, and partially used study drugs at the next visit. The patient will be instructed to take the pre-specified number of tablets of the study drug by mouth two times daily starting in the evening after this Visit. The evening dose should be approximately 12 hours after the morning dose. Document that the patient understood the dosing instructions.

The patient will leave the clinic with enough IMP for the next 3 months  $\pm$  7 days and begin to take the assigned IMP (nabilone) in the evening after this visit.

#### 5.5 Termination Visit / V 3

After 6 months of open-label nabilone treatment, the patient will return to the clinic to perform his/her termination Visit / V3. The time and date of the last dose of study drug will be

documented.

The following assessments should be performed and documented with date and time at this visit:

- 1. Perform assessment of Vital signs: obtain weight, temperature, obtain and record serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing
- 2. Ask for AE occurring since the last visit.
- 3. Interview on concomitant medication use since the last visit.
- 4. Perform physical and neurological examination
- 5. Urine sample for pregnancy test (for women of childbearing potential only)
- 6. Administer the MDS-UPDRS Part I, II, III, and IV (record if patient is in ON or OFF state), and the Modified Hoehn and Yahr stage
- 7. Administer the following assessments:
  - a. NMSS
  - b. HADS
  - c. PDQ-8
  - d. ESS
  - e. FSS
  - f. KPPS
  - g. CGI-I
  - h. C-SSRS
  - i. QUIP-RS
  - j. MoCA
  - k. MMSE
- 8. Collect all used, unused, and partially used study drug and record it in the source documents and Drug Accountability Section.

Nabilone will then be down-titrated in 0.25 mg decrements every other day until it is discontinued. During dose tapering phone calls will be held every other day to receive information on AEs, Concomitant Medication use, CGI-I, the items 1.2, 1.8, and 1.12 of MDS-UPDRS Part I, and the C-SSRS will be executed. A phone call for safety issues will be held after 5 days  $\pm$  2 days and a Safety Follow- Up Visit will be scheduled after 2 weeks + 2 days of discontinuation from study drug. (see 5.6)

The Safety Follow- Up Visit should be scheduled with the patient and he/she should be reminded on the telephone calls. Relevant contact to the site should be updated if necessary if there are any questions or adverse events occurring until the Safety Telephone Call or Follow-Up Visit.

## 5.6 Safety Telephone Call (TC – S) and Safety Follow-Up Visit (V – S)

The **Safety Telephone Call** will be held after 5 days  $\pm$  2 days after stopping the study drug and will include the assessment of AE, concomitant medication, and the CGI-I.

Questions for the following items and assessment of the following scale will be performed:

- Hallucination item (1.2) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society –
   Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Day-time sleepiness item (1.8) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- C-SSRS

Documentation in the source document will include the time and date of the call as well as the results of the assessments.

The **Safety Follow-Up Visit** will take place 2 weeks + 2 days after the withdrawal from study drug and will include the following assessments (documented with date and time in the source documents):

- 1. Perform assessment of Vital signs: obtain weight, temperature, obtain and record serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing
- 2. Ask for AE occurring since the discontinuation of the study drug.
- 3. Interview on concomitant medication use since the last intake of study medication.
- 4. Perform physical and neurological examination
- 5. Administer the MDS-UPDRS Part I, II, III, and IV and the C-SSRS and the CGI-I
- 6. Collect all used, unused, and partially used study drug and record it in the source documents and Drug Accountability Section.

#### 5.7 Early Termination Visit

If the patient has discontinued the IMP prematurely, an early termination visit should be performed as soon as possible after the last dose of study drug and the Sponsor should be informed. The date of the last intake of study drug should be documented and a reason for withdrawal of the study drug if available. This visit will include the following assessments (documented with date and time in the source documents):

1. Perform assessment of Vital signs: obtain weight, temperature, obtain and record

serial BP and pulse measurements after at least 10 minutes of supine rest and again after 1, 3, 5, and 10 minutes of active standing

- 2. Ask for AE occurring since the discontinuation of the study drug.
- 3. Interview on concomitant medication use since the last intake of study medication.
- 4. Perform physical and neurological examination
- 5. Urine sample for pregnancy test (for women of childbearing potential only)
- 6. Administer the MDS-UPDRS Part I, II, III, and IV (record if patient is in ON or OFF state), and the Modified Hoehn and Yahr stage
- 7. Administer the following assessments:
  - a. NMSS
  - b. HADS
  - c. PDQ-8
  - d. ESS
  - e. FSS
  - f. KPPS
  - g. CGI-I
  - h. C-SSRS
  - i. QUIP-RS
  - j. MoCA
  - k. MMSE
  - Eye-tracking (only to be performed if ET is performed before V 2)
- 8. Collect all used, unused and partially used study drug kits and document in the source documents and Drug Accountability Section.

A Safety Follow-Up Visit should be performed 2 weeks + 2 days after the last intake of study medication (if the Early Termination Visit occurs not longer than 5 days after the discontinuation of the study medication).

#### 5.8 Unscheduled Visit / USV

An Unscheduled Visit is defined as any additional visit performed at any time between the Screening / Baseline Visit and the Safety Follow-Up Visit. This visits can be held at the investigator's

discretion. An USV should at least contain questions and assessments for:

- 1. AE occurring since the last visit.
- 2. Concomitant medication use since the last visit.
- 3. CGI I
- 4. C-SSRS
- 5. Obtain and record the date and approximate time when the patient took the most

recent dose of IMP. Collect all used, unused, and partially used study drug kits dispensed at the previous visit and document in the source documents and Drug Accountability Section. Assess compliance. Document any missed doses, lost tablets, and number of tablets taken

The reason for the Unscheduled Visit should be provided and recorded in the source documents. Additional assessments can be performed if necessary by the means of the investigator including a neurological and physical exam, a pregnancy test, and the clinical scores used in the trial.

#### 5.9 Telephone calls

Telephone calls will be performed according to the study protocol during the dose titration phase and during dose tapering as summarized in 3.2 (Schedule of Events). Telephone calls will be held every other day (1) during dose titration phase until optimal dose will be reached and (2) during dose tapering until IMP is stopped. A Safety Telephone Call will be held 5 days  $\pm$  2 days after discontinuation of study medication. During these telephone calls patients will be asked for any AEs, SAEs, and the CGI-I. Moreover, the hallucination item (1.2), the day-time sleepiness item (1.8), the OH item (1.12) of the MDS-UPDRS, and the C-SSRS will be applied.

If the site is not able to reach a patient (or study partner) via telephone on the scheduled day and all attempts have been made and there is no other possibility to reach the patient and no reasonable explanation, the site is allowed to stop trying to connect to the patient. At least 3 attempts have to be made. Attempts have to be documented as well as the decision to discontinue trying. The site has to attempt to reach the patient on the consecutive working day again.

If a telephone call is scheduled on a Saturday, the patient should be reached on Friday. If a telephone call should be held on Sunday, the call will be scheduled on Monday. On bank holiday, the patient should be called the day before or after the day off.

The patients will be provided with an emergency phone number available 24 hours to contact a member of the study team in case of emergencies.

# 6 Description of Assessments: Efficacy and Safety Variables

#### 6.1 Secondary Endpoints: Assessments of Efficacy

The secondary endpoints will be measured as the change in the clinical scales and questionnaires regarding motor symptoms and different domains of non-motor symptoms in Parkinson's Disease between V 1 and the termination visit. For the MoCa and the MMSE, the difference between the Screening Visit of the NMS- Nab Study and the Termination Visit of this extension study will be compared.

Therefore, the total MDS-UPDRS Part I, II, III, and IV (total UPDRS: 50 items, Part I: 0 to 52 points, Part II: 0 – 52 points, Part III: 0 – 132 points plus Hoehn and Yahr Scale 0 - 5 points, Part IV: 0-24 points), the Non Motor Symptoms Scale (4 domains, 15 items, points from 0 – 12x15 with the latter being severely impaired daily or always), the Hospital Anxiety and Depression Scale (14 items, values from 0 – 42 points), the Parkinson's Disease Questionnaire – 8 (8 items), the Montreal Cognitive Assessment (8 items, score ranges from 0 – 30 points), the Mini Mental State Exam (0 to 30 points), the Epworth Sleepiness Scale (8 items, ranges from 0 – 24 points), the Fatigue Severity Scale (9 items, 9 – 63 points), the King's Parkinson's Disease Pain Scale (7 domains, 14 items, 0 – 168 points), and the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease–Rating Scale (7 domains, 0 – 122 points) will be performed. The result of the Clinical Global Impression – Global Improvement scale (ratings from 1 to 7) at the Termination Visit will be used as a secondary efficacy criterion. All presented scales are measured in points given above.

Currently, the MDS-UPDRS Scale is the most common used scale in evaluation motor symptoms in patients with PD. The Movement Disorder Society (MDS)-sponsored new version of the UPDRS was published in 2003 with respect to the Task Force for Rating Scales' proposed criticism of the original UPDRS concerning issues of weakness and ambiguities. (44) The scale consists of four components with each part addressing different domains of symptoms of PD and its therapy (Part I: Non-Motor Experiences of Daily living; Part II: Motor experiences of daily living; Part III: Motor Examination; Part IV: Motor Complications). Each section was written by appropriate members of the subcommittees, reviewed, and ratified by the subcommittee. Part I of the MDS-sponsored new version of the UPDRS consists of one part (Part IA) containing the observations of the investigator regarding behaviors based on information from patients and caregivers, and one part (Part IB) to be self-administered by the patient alone or with help of the caregiver without

cooperation with the investigator. The rater can solely review this part to ensure that all items are rated and questions for understanding can be addressed to him/her. Part II is also based on the patient's self-evaluation. Part III needs to be demonstrated or performed by the rater. Part IV consists of instructions for the investigator and the patients to combine clinical observations with information provided by the patient and it is executed by the rater. Only qualified and trained raters will administer the MDS UPDRS subscales in accordance with requirements for background and experience in research settings. Trainings will be documented by providing a Certificate of Rater Approval. The MDS UPDRS Scale will first be measured before the patient receives nabilone and in subsequent visits after the patient's morning dose of nabilone. It will be documented if the patient is in an ON state (i.e. period when the patient notices a benefit on MS from standard oral LD/CD treatment) or in an OFF state (i.e. the phase with no response to medication and significant motor symptoms).

The **Non-Motor Symptoms Scale (NMSS)** was developed by an international multidisciplinary PD-NMS group in order to create a comprehensive questionnaire to assess symptoms of PD that are not affecting movement. Symptoms included in the scale range from vertigo and other symptoms of orthostatic hypotension, falls, daytime sleepiness and subsequent loss of energy, sleep disturbances at night, restlessness in the legs to psychiatric and cognitive symptoms like apathy, loss of motivation and interest, nervousness, anxiety, worry, sadness, depression, mood swings, loss of joy in usual activities, and symptoms of delusion, hallucinations, and double vision.

The **Hospital Anxiety and Depression Scale** was developed in 1983 from Ziegmond und Snaith which edited a longer version of the questionnaire and published this 14-items-long tool. The Scale aims to assess symptoms of anxiety and depression and was generated as a screening tool. 7 items address symptoms of anxiety and the other 7 items assess depression in patients. Therefore, a subscore for anxiety and depression can be generated. Questions regarding physical symptoms and intrusive items are not included to avoid confounding of the result by organic diseases.

#### Parkinson's Disease Questionnaire-8

The PDQ-8 is the short version of the longer PDQ-39 scale and was created to measure the health status and functional capacity of patients with PD. Its eight questions cover eight aspects of quality of life. The instrument was developed on the basis of interviews with people diagnosed with PD and it has been widely validated. The questions relate to mobility, activities of daily living, emotional well-being, social support, cognition, communication, and

bodily discomfort. The patient is asked to rate each question regarding his/her PD symptoms over the past month.

#### **Montreal Cognitive Assessment Scale (MoCA)**

Nasreddine et. al created the MoCA in 1996 in Montreal, Quebec to asses symptoms of mild cognitive impairment. The test assesses several cognitive domains through its task for orientation to time and place (6 points), its learning task (five nouns) to assess short-term memory recall (5 points), a task to assess visuospatial / executive functions (task adapted from trail making B task, clock-drawing task, and drawing a three-dimensional cube, 5 points), and a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points).

Cognitive function and working memory are evaluated using a sustained attention task (target detection using tapping,1 point), a serial number subtraction task (3 points), and a task where digits are repeated forwards and backwards (1 point each). Verbal skills are assessed by using a confrontation naming task with animals with low familiarity (lion, camel, rhinocerus, 3 points), by letting the patient repeat two sentences with complex syntax (2 points), and the fluency task described above.

#### Mini Mental State Exam (MMSE)

Folstein et al. developed the MMSE in 1975. The MMSE is a The MMSE consists of 30-items and was designed to be a brief global cognitive screening measure. It consists of several short tasks used to assess attention, memory, language, and visuospatial abilities, as well as orientation to person, place and time. A cutoff of 24 (23 and below) has been proposed to detect cognitive impairment.

#### **Epworth Sleepiness Scale (ESS)**

Daytime sleepiness is assessed by the ESS, which is a short self-administered scale asking for the probability of dozing in eight different situations during the day. Answers can range from no chance of dozing to high chance of dozing in the following scenarios: sitting and reading, watching TV, sitting in a public space, being an assistant driver in a one-hour ride without a break, relaxing in the evening, sitting and talking to another person, sitting still after lunch without intake of alcohol and stopping the car at a traffic light.

#### King's Parkinson's disease pain scale (KPPS)

Chaudhuri et al. initially published the KPPS to be a reliable and valid scale to rate different types of pain in PD in 2015. (45) Its aim is to evaluate the global and bedside burden of pain and to characterize various phenotypes of pain in Parkinson Disease (PD) patients.

The scale consists of seven domains including 14 items, with each item scored by severity (0-3) multiplied by frequency (0-4), resulting in a subscore of 0 to 12, with a total possible score range from 0 to 168. The KPPS provides questions for musculoskeletal pain, chronic pain, fluctuation-related pain, nocturnal pain, oro-facial pain, discolouration, oedema / swelling and radicular pain.

The contact information for this questionnaire and the permission to use for this study was granted by: Mapi Research Trust, Lyon, France – Internet: https://eprovide.mapi-trust.org

#### **Fatigue Severity Scale (FSS)**

To evaluate the level and severity of fatigue of patients during the past week the FSS will be used in this study. It consists of nine statements with levels ranging from 0 to 7 points whereat a low value indicates a strong disagreement with the statement and a high value a strong approval of it. The scale pays attention to motivation, the impact of exercise on fatigue, the impact of fatigue on (physical) functioning, work, family or social life, and problems and disability arising from fatigue.

#### Clinical Global Impression - Improvement (CGI-I)

The CGI-I is used by the investigator to rate the patient's total improvement based on a 1 to 7 point weighted scale at which one point means "very much improved" and seven points indicate a status of being "very much worse". If the scale has not been assessed, a zero score will be given. The rater should evaluate the improvement of the patient to his clinical judgment, whether or not the improvement is believed to be due to drug therapy.

### Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS)

The QUIP-RS is a measurement designed to support the diagnosis and to measure the severity of symptoms of impulse control disorders and related disorders in PD in the last four weeks. The QUIP-RS consists of 4 primary questions addressed to commonly reported thoughts, urges/desires, and behaviours associated with impulse control disorders each applied to 4 domains of impulse control disorders and 3 domains of related disorders. These 4 domains are: compulsive gambling, buying, eating, and sexual behavior. The 3 domains of related disorders are medication use, punding, and hobbyism. Each question can have a score from 0 to 4 assessing the frequency of thoughts, urges, or behaviours. The scores for each impulse control disorder and related disease can range from 0 to 16 points, with a higher score indicating a greater severity of symptoms. The total QUIP-RS score for all ICDs and related disorders combined can have values from 0 to 112 points.

© University of Pensylvannia

#### 6.2 Primary Endpoints: Safety Assessments

The primary endpoint of this study is to evaluate long-term (from V 1 Visit to the Termination Visit) safety and tolerability of nabilone for non-motor symptoms in PD patients.

#### **Tolerability** will be described through the:

- Number of subjects (%) who discontinue the study
- Number of subjects (%) who discontinue the study due to AE

#### Safety Measures include the following:

- Adverse Events (AE), Serious Adverse Events (SAEs), Suspected Unexpected Serious Adverse Reactions (SUSARs)
- Clinical assessment
- Vital signs including performance of active orthostatism (measurement of heart rate and blood pressure after 10 minutes of quiet rest in the supine position and at 1, 2, 3, 5, and 10 minutes of active standing)
- Patient's Compliance
- Prior and Concomitant Medication Use
- Hallucination item (1.2) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Orthostatic hypotension (OH) item (1.12) of Movement Disorders Society –
   Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Day-time sleepiness item (1.8) of Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Columbia Suicide Severity Rating Scale (C-SSRS)

## 6.2.1 Adverse Events, Serious Adverse Events, Adverse Drug Reaction, Suspected unexpected serious adverse reactions

Safety assessment can be implemented by monitoring and recording of AEs including ADR, SAEs, and SUSARs. For a description of the terms, documentation, and reporting see 8 of this protocol. The patients should be questioned for adverse reactions at any visit and telephone call. This should be reported on the CRF and in the patient's record. In case of an SAE or SUSAR, an immediate (within 24 hours) reporting to the Sponsor and the competent authorities is obligatory.

#### 6.2.2 Description of other safety measures

#### **Demographics**

At the Screening / Baseline Visit, the patient will be asked for ethnicity, sex, age at examination, year and age of symptom onset, marital state, education (years), profession, family history (brief), and social history (brief).

#### Physical and neurological examination

A brief physical and neurological examination of the patient will be held at the Screening / Baseline Visit, the Visits V 1, V 2, V 3, the Safety Follow-up Visit, and an Early Termination Visit (if applicable) of the patient and documented in the patient's record.

All physical examinations will be performed by trained medical personnel only, prior to IMP administration on dosing days. Any abnormal findings will be recorded as AEs.

Physical examination must at least include assessment of the vigilance and orientation, general condition, nutritional condition, HEENT (head, eyes, ears, nose and throat), respiratory system, heart, abdomen, extremities, and visible skin and mucous membrane. Patients should be guestioned for defecation and the act of urination.

Neurological examination should include standard neurological assessment of vigilance, orientation, mental status (e.g. consciousness), meningism, cranial nerves, the motor system and sensory system of both upper and lower extremities, reflexes (including pathological reflexes), cerebellar signs, gait, tandem gait, and postural stability, as well as special tests for parkinsonism (e.g. finger tapping, toe tapping, facial expression, ...).

#### Vital signs

Vital signs including the evaluation of weight, height (only at Screening / Baseline Visit), temperature, and active orthostatism will be performed at all visits during the course of the study. The latter will be assessed by measuring the heart rate and blood pressure after 10 minutes of quiet rest in a supine position and at 1, 2, 3, 5, and 10 min after active standing. Blood pressure and pulse rate should be obtained in a quiet room at a comfortable temperature, with the patient's arm unconstrained by clothing or other material, and with an appropriate cuff size. In this study, an automatic BP cuff (sphygmomanometer) with digital advert will be used. Patients with symptomatic orthostatic hypotension will be excluded from the study.

#### **Concomitant medications**

The patients will be asked for concomitant medication on every visit and telephone call and will be assessed in regard to permitted and prohibited concomitant medication.

#### **Patient's Compliance**

The patient's compliance will be assessed by open questions from the investigator at every on-site visit and phone call.

# Hallucination item (1.2) of MDS-UPDRS Day-time sleepiness item (1.8) of MDS-UPDRS Orthostatic hypotension (OH) item (1.12) of MDS-UPDRS

These items are part of the UPDRS Part I (Mental Activity, Behaviour, and Mood) and refer to delusions and hallucinations of all sensations and to the loss of insight of the patient, to day-time sleepiness and its frequency while reading or watching TV, while having a discussion or during the meal, and to the sensation of drowsiness and vertigo and its consequences, like falls during the last week.

The items are assessed to detect potential side effects that may occur due to drug treatment. The will be assessed at every clinical visit and during all phone calls and documented in the source documents.

#### **Columbia Suicide Severity Scale (C-SSRS)**

The C-SSRS was initially designed for suicidal assessment in one study, but has shown overall successful prediction of suicidal behaviour in adolescences and adults. It is the only screening tool to assess the full range of suicidal ideation and behaviour including criteria for the next steps (e.g. referral to a mental health professional). Suicidality in this study with this scale will be assessed by trained study personnel only (Posner et. al, 2011) on all visits and telephone calls as a measurement for safety. The scale consists of 4 categories: suicidal ideation, intensity of suicidal ideation, suicidal behaviour, and actual/potential lethality which can be answered by Yes or No. At Screening / Baseline Visit the questionnaire for the past 6 months will be used and for all other visits and phone calls the version "Since the last visit" will be administered.

© 2008 The Research Foundation for Mental Hygiene, Inc.

#### 6.3 Assessment of exploratory endpoint

Eye-tracking Examination (reaction time, attention span, concentrativeness)

#### Eye-tracking: Measurement of eye-movements with the Tobii TX-300

Eye-tracking provides a fast and non-invasive method for various examinations. In this study we will measure the reaction time using prosaccade and antisaccade tasks. Moreover, we will assess attention spans and the concentrativeness using a customized saccade task and a test involving task-switching. The examination will be performed at the Visit V 2. Examinations will take place in a quiet room by trained personnel only.

#### 7 Study Treatments

#### 7.1 Details of Study Treatment

## 7.1.1 Name and Description of Investigational Medicinal Product (IMP) and Comparator

#### Nabilone:

Nabilone is a synthetic cannabinoid derivative. Canemes 0.25 mg capsules are an oral dosage form in white hard gelatine capsules. Each capsule contains 0.25 mg Nabilone as the active ingredient, in the form of a polyvinylpyrollidone (Povidone) co-precipitate and corn starch. Each PE bottle contains 28 capsules for a treatment period of approximately 1 month.

Synthetic cannabinoid nabilone

Other components: Polyvinylpyrollidone (Povidone) co-precipitate and corn starch

Administration form: capsules

Mode of administration: oral

Dose: 0.25 - 2 mg per day

Manufactured in 0.25 mg dosage strength

Bottles of 28 capsules each

For clinical trial use only, Usage as described in the protocol

Stored at room temperature,

Store pharmaceutical material out of the reach and sight of children

Sponsor: Medical University of Innsbruck, Austria

Represented by O.Univ.-Prof. Dr. Werner Poewe

#### 7.1.2 Dosing Instructions

During titration phases nabilone will be started with a dosage of 0.25 mg in the evening orally and titrated by 0.25 mg increments every one- to four- daily. Dose adjustments should be performed as follows:

First dose to be implemented: 0.25 mg orally in the evening once a day (0-0-1)

Increase in one to four-day- steps, according to the investigator's decision:

- 2. 0.25 mg by mouth BID (1-0-1),
- 3. 0.25 mg 1-0-2 orally,
- 4. 0.25 mg 2-0-2 orally,
- 5. 0.25 mg 2-0-3 by mouth,
- 6. 0.25 mg 3-0-3 orally,
- 7. 0.25 mg 3-0-4 p.o.,
- 8. 0.25 mg 4-0-4 orally

A maximum of 1 mg twice a day should not be exceeded. Optimally, the dose the patient was classified as a responder in the NMS-Nab Study should be reached. However, the

investigator can adapt this dose according to his/her decision. Between morning dose an evening dose a time interval of 12 h should be meet. Preferably, tablets should be taken at the same time each day. In case a participant misses a dose, he/she will be instructed to take their next dose of nabilone at the normally scheduled time.

The increment of dosage should take place until the patient has much (CGI- I Rating Scale: 2) or very much (CGI-I Rating Scale: 1) improved, reached a maximum dose of 1 mg BID or experiences intolerable adverse events that are believed to be related to the study drug.

During the trial the fixed dosage of the study drug should not be changed. If the patient deteriorates in his CGI-I, dose adjustments can be made and the patients doesn't have to restarts again at titration phase.

#### 7.1.3 Packaging and Labelling

The IMP supplies for this study will be packaged according to current GMP guidelines and applicable national laws and regulations. For titration phase, IMP will be packaged in an open-label fashion. Packaging, labelling and distribution of IMP will be performed by the company Kwizda.

#### 7.1.4 Handling and Storage Requirements

The investigators will be responsible for ensuring the correct storage and sufficient stocks of the IMP and comparative drug at the trial centers. The investigator bears the responsibility for the proper storage in a secure location at the site which means in a lockable cabinet with restricted access to the investigator(s) and authorized site staff. Personnel having access to the IMP will be listed on the Authorization and Delegation log in the Investigator Site File (ISF). The investigators will ensure that the IMP is only used according to this protocol and will only be dispensed to participants of the study. Dispensing will be performed by authorized members of the study team. The investigator will be responsible for the Drug Accountability log. Drug accountability will be recorded in the patient's record as well. Drug accountability will be noted by a monitor during site visits and at the completion of the trial. Unused study drug from all sites will be sent to the company Kwizda for destruction after completion of the trial (LPLV).

#### 7.2 Subject's Compliance

#### 7.2.1 Numbering of Patients

All participants who are eligible for the study (see: Inclusion criteria 4.1.) will receive a

continuous number according to their enrollment in the study.

This will be a unique number received at the Screening / Baseline Visit to be identified throughout the participation in the study (in ascending order, starting with number 001 for the first patient). This number will be used in all communications between the investigator and the Sponsor for the specific patient. A patient only enters the trial, if he meets all inclusion and none of the exclusion criteria during the Screening / Baseline Visit. The assigned kit number of the open-label IMP will be documented in the source documents.

In case of a drop-out, no replacement will be recruited and the screening number will be assigned as before in an ascending order.

Due to this study being an open-label study, no procedures for blinding and unblinding are outlined in this protocol.

#### 7.3 Drug Accountability and Treatment Compliance

The receipt of medication and the condition of it as well as the loss or damage of medication will be recorded in the source documents and the company Kwizda will be informed. The dispensing and return of medication should be documented in the Drug Accountability Section and the patient's record. Both this records and the medication supplies must be available to be reviewed by the study Sponsor or designee at any time requested. The investigator is responsible for appropriate storage of used, unused, and partially used study drug supplies on-site until they are returned for destruction on completion of the study (LPLV).

Supplies of nabilone intended for this study should only be used for the purpose of the study and adhering to this protocol. It is prohibited to apply for any other purpose. The investigator is responsible that the use of the study drug is strictly in accordance with the study protocol.

#### 7.3.1 Procedures for Monitoring Patient Compliance

In outpatient treatment procedures for the verification and documentation of the compliance will be as follows:

- The patients only receive the amount of medication units at each visit that will be needed until the next visit.
- The Investigator takes back the empty containers or non-used units.

The patient must return all used, unused, and partially used study drug supplies at the planned visits in the study course. Drug accountability must be done in the presence of the participant. Thus, discrepancies between the dosing regime and the patient's compliance
can be clarified directly. Drug Accountability must be recorded in the source documents and the Drug Accountability Log in the Investigator Site File.

The end of treatment for the patient should be documented.

In case of persistent noncompliance of a patient (<80% to >120% of the assigned dose), the Sponsor or its designee will be informed to decide together with the investigator whether the patient should be discontinued or not.

#### 7.4 Prior and Concomitant Medications/Treatments

#### 7.4.1 Allowed Anti-PD Medications/Treatments

All Anti-PD Medications are allowed in this study preconditioned the patient has a stable Parkinson's disease and that the regimens of Anti-Parkinson's medications, other current prescribed/non-prescribed medications or dietary supplements are stable for at least 30 days prior to screening and will be continued on the same doses and regimens. The nabilone titration in the NMS-Nab Study should be an exception of this.

The addition of any new anti-PD medication or other prescribed / non-prescribed drugs are allowed during the study as well as changes to frequency or intervals between doses, but have to be recorded in the source documents and discussed with the investigator due to possible interactions.

Participants will be advised to refrain from the use of any concomitant medication during their participation in the study without prior permission by the investigator. The use and the reason for the use of any additional medication will be recorded in source documents.

#### 7.4.2 Prohibited Concomitant Medications/Treatments

Nabilone has an addictive and CNS depressing effect if taken together with diazepam, Na-Secobarbital, alcohol and codeine.

Interactions between nabilone and the following medications have been observed. Therefore, these the intake of these drugs during the course of the clinical trial is prohibited for participants of this study.

- amphetamine, cocaine, other sympathomimetics
- atropine, scopolamine, antihistaminics, other anticholinergic substances
- amitriptyline, amoxapine, desipramine, other tricyclic antidepressive drugs
- barbiturates, benzodiazepines (except for clonazepam up to a maximum of 1.5 mg per d), lithium, opioids, buspirone, muscle relaxing agents, CNS depressing substances
- disulfiram

- fluoxetine
- antipyrines
- theophylline
- naltrexone

# 7.5 Concomitant Non-Pharmacologic Therapies

All non-pharmacological therapies (physical therapy, exercise, yoga, ...) the patient performs to improve his/her parkinson symptoms can be continued during participation in the study. During the trial, such non-pharmacological therapies can be started as well. All non-pharmacological therapies will be documented in the source documents at the Screening / Baseline Visit. The concomitant non-pharmacological therapies should be kept on the same levels during the study.

#### 8 Adverse Events

# 8.1 Summary of known and possible Adverse Events of the IMP

Generally, nabilone is well tolerated.

Common adverse reactions (>1/100 to <1/10) observed in patients are:

- Somnolence
- Vertigo
- Euphoria
- Ataxia
- · impaired vision
- difficulties to concentrate
- sleep disturbances
- dysphoria
- headache
- hypotension
- nausea
- dry mouth

Controlled trials with patients taking nabilone showed that at least one side effect occurred per subject. Most patients develop a tolerance in regard of adverse events concerning the CNS and therefore relaxation, somnolence and euphoria reside after some weeks. This effect is reversible.

In therapeutic doses nabilone is a potential addictive drug. The potential to cause mental addiction is unknown and no patient has shown withdrawal symptoms in clinical trials. In conjunction with psychological stress, an **overdose phenomenon** of nabilone can appear at therapeutic doses. Symptoms due to overdosing nabilone have been described as enhanced psychomimetic and psychological side effects of the drug. In clinical trials a normalization of the mental state of the patient was reached after 72 hours of withdrawal of the drug without additional therapy. One should monitor vital signs due to the possible occurrence of hypertension, hypotonia, and tachycardia.

No cases of patients taking doses above a level of 10mg daily have been described in clinical trials so far. Hereby, one would expect symptoms like hallucinations, anxiety, respiratory depression, and coma.

No adaption of dose needs to be done in the elderly. Nabilone should not be used in patients under the age of 18 years because it has not been studied in separate trials. The primary route of elimination of nabilone is biliary. Thus it should not be used in patients with severe impairment of liver function. No data in patients with impaired renal function have been collected, which is why it should be used with caution in these patients.

**Nabilone should not be used during pregnancy or lactation** because of the lack of data in this cohort. In experiments with animals, no reproductive toxicity has been described. No studies on carcinogenesis have been performed.

#### Minor risks of nabilone (>1/10.000 to <1/1.000) include:

- Confusion
- Disorientation
- Hallucination
- Psychosis
- Depression
- difficulties in coordination
- tremor
- loss of appetite
- anxiety
- depersonalisation
- tachycardia
- abdominal pain

The IMP can cause alterations of physical and mental capabilities which are essential for tasks requiring high attention e.g. driving or operating machines. The study medication can be detected in the body after withdrawal (total half-life 35 hours) which could lead to misinterpretation in case of a control through regulatory authorities e.g. police.

## 8.2 Definition of an Adverse Event (AE)

An adverse event is "any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment". (47)

An AE can therefore be any unfavourable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease which is considered to be clinically relevant by the physician and is temporally associated with the use of a medicinal

(investigational) product, whether or not related to the study drug.

Adverse events include:

- Worsening or increase in frequency or intensity of a pre-existing disease or medical condition in an unexpected manner
- Abnormal laboratory tests (clinically significant)

#### Adverse events do not include:

- Pre-planned interventions/hospitalizations
- Medical or surgical procedures, e.g. surgery, endoscopy, tooth extraction, transfusion. However, the event leading to the procedure is an AE. If this event is serious, the procedure must be described in the SAE narrative.
- Pre-existing disease or medical condition that does not worsen.
- Overdose of either study drug or concomitant medication without any signs or symptoms.

In order to ensure complete safety data collection, all AEs occurring during the study (i.e., after the signing of the ICF), including any post-treatment periods required by the protocol, must be recorded in source documents even if no investigational product was taken but specific study procedures were conducted. This includes all AEs not present prior to the Screening / Baseline Visit and all AEs that occurred or worsened after the Screening / Baseline Visit. Events that occur prior to giving informed consent are captured as medical history.

Signs or symptoms of the disease for which the investigational product is being studied should be recorded as an AE if their frequency or intensity increases in a clinically significant manner or their nature changes unexpectedly as compared to the clinical course known to the investigator from the patient's history, or the natural course of the disease.

## 8.3 Definition of a Serious Adverse Events (SAEs)

"A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect". (47)

An adverse event is therefore considered serious by the definition by the International Conference on Harmonization (ICH) guidelines if it can be characterized by at least one of the following criteria:

Results in death

- is life-threatening defined as an event in which the subject was, in the judgment of the investigator, at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it had been more severe.
- requires inpatient hospitalization or prolongs an existing hospitalization
- causes persistent or significant disability or incapacity (i.e. a substantial disruption of a person's ability to conduct normal life functions)
- or is a congenital anomaly/birth defect (including that occurring in a fetus)
- or requires medical or surgical intervention to prevent one of the above mentioned outcomes. (i.e. the development of drug dependency or drug abuse)

Inpatient hospitalization is defined as an overnight stay in a hospital unit and/or emergency room that includes at least one night (midnight to 06:00 AM).

The following is not considered as a SAE and should be reported as an AE only:

 Treatment of an emergency or outpatient basis for an event not fulfilling the definition of seriousness given above and not resulting in hospitalization

The following reasons for hospitalization are not considered as AEs or SAEs:

- Standard monitoring of a pre-existing disease or medical condition that did not worsen, e.g. hospitalization for coronary angiography in a subject with stable angina pectoris
- Elective treatment of a pre-existing disease or medical condition that did not worsen, e.g. hospitalization for chemotherapy for cancer, elective hip replacement for arthritis
- Hospitalization for cosmetic elective surgery, social and/or convenience reasons

A change in vital signs, diagnostic tests (e.g., an electrocardiogram), or laboratory test results may be an SAE if the change meets one of the above criteria.

# 8.4 Adverse Drug Reaction (ADR) & Unexpected Adverse Drug Reaction

An ADR is any noxious and unintended response to an IMP related to any dose with at least a reasonably possible causal relationship with the IMP.

Unexpected ADR means the nature or severity of which is not consistent with the applicable product information available for the IMP. Expected ADRs are listed in the appropriate reference documents (e.g. Investigator's Brochure).

# 8.5 Suspected Unexpected Serious Adverse Reactions (SUSARs)

A SUSAR is an event that is believed to be at least possible related to the administration of the study drug and is severe and unexpected. It therefore may illustrate a side effect of the drug. For clinical studies in which an IMP is used, the FDA defines an "unexpected" AE as an AE that has never been seen before, or is not consistent with the information about the drug's risks in the relevant source documents (e.g. Investigator's Brochure).

# 8.6 Pregnancy

In the event a patient becomes pregnant after the first intake of any IMP, the investigator and the Sponsor should be informed immediately. The patient should be withdrawn from the study as soon as pregnancy is known, and should immediately stop the intake of the IMP. If a pregnancy should be confirmed after informed consent has been obtained but prior to the initiation of the study drug, the patient must be excluded from the trial. The pregnancy must be followed up to determine outcome (including premature termination) and status of mother and child. Pregnancy complications (including spontaneous abortions) and elective terminations must be reported as an AE or SAE. Any SAE occurring in association with a pregnancy brought to the investigator's attention after the subject has completed the study and considered by the investigator as possibly related to the IMP, must be promptly reported to the Sponsor.

The participant should return for an Early Termination visit as soon as possible and should be followed by via a Safety Follow-Up Visit 14 days + 2 days after discontinuation of the study drug (if the ET is performed after 5 days after the last intake of study drug). The investigator must inform the patient of currently known potential risks for pregnancy outcome and available treatment alternatives.

In case the partner of a male patient enrolled in the clinical study becomes pregnant, the Sponsor must be informed immediately by the investigator or designee and a decision of the further procedure will be made.

The pregnancy will be documented in the source documents including the progression of the pregnancy and the eventual date of birth (if applicable) as well as the health of the mother and of the child. The health of the child must be followed for 30 days after birth for any significant medical issues.

A pregnancy becomes an SAE in the following circumstances: miscarriage, abortion, or anomaly/birth defect of the child. Those SAEs must be reported to the Sponsor as described below.

As the consent for the study does not cover the consent for the follow-up of the pregnancy, a separate consent has to be obtained.

## 8.7 Overdose of Investigational Medicinal Product

If the patient has taken a dose beyond that prescribed in the protocol (including section on overdose) should be recorded in the source documents and in the Drug Accountability. These events are only considered to be AEs or SAE if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (e.g., suicide attempt). Any SAE or nonserious AE associated with excessive dosing must be followed as any other SAE or AE.

## 8.8 Grading of Severity of Adverse Events

The term "serious" in SAE refers to the outcome of a patient's event that poses a threat to his/her life or functioning rather than to its intensity, which is described by the term "severity". In the latter, the event itself may be of relatively minor medical significance (such as a severe headache).

Intensity of all adverse events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03 on a five-point scale (grade 1 to 5) and reported in detail in the patient's records and CRF.

Adverse events not listed in the CTCAE version 4.03 should be graded as follows:

Table 4: CTC grading of Adverse Events

| CTC grade | Equivalent to | Definition |
|---|---|---|
| Grade 1 | mild | Discomfort noticed but no disruption of normal daily activity |
| Grade 2 | moderate | Discomfort sufficient to reduce or affect daily activity; no treatment |
| | | or medical intervention is indicated although this could improve the |
| | | overall wellbeing or symptoms of the patient. |
| Grade 3 | severe | Inability to work or perform normal daily activity; treatment or |
| | | medical intervention is indicated in order to improve the overall |
| | | wellbeing or symptoms; delaying the onset of treatment is not |
| | | putting the survival of the patient at direct risk. |
| Grade 4 | | An immediate threat to life or leading to a permanent mental or |
| | life-threatening | physical condition that prevents work or performing normal daily |
| | / disabling | activities; treatment or medical intervention is required in order to |
| | | maintain survival. |

| Grade 5 | death | AE resulting in death |
|---------|-------|-----------------------|

## 8.9 Causality

The assessment of relationship of adverse events to the administration of IMP is a clinical decision based on all available information and considering all relevant factors such as (but not limited to) the underlying indication, coexisting diseases, concomitant medication, etc. at the time of the completion of the patient's record and case report form of this visit.

The term "related" refers to the ability of the study drug to cause the AE implicating a relationship in time and that the event would not have happened without the effort of the study drug.

The question: "Is there a reasonable possibility that the study drug caused the event?", should be asked. Answer **YES** (possibly, probably or definitely related) if one or more of the following criteria apply:

- The event follows a reasonable temporal sequence from administration of study drug
- The event could not be reasonably attributed to the known characteristics of the patient's clinical state, environmental or toxic factors or other modes of therapy administered to the patient
- The event follows a known pattern of response to study drug
- The event disappears or decreases on cessation or reduction in dose of the study drug. (It should be noted that in some situations an AE will not disappear or decrease in intensity upon discontinuation of study drug despite other clear indications of relatedness).

Otherwise answer **NO** (not related).

Moreover, the relationship between the AE and the study drug can be described stepwise:

- definitely related: an AE that follows a temporal relationship with implementing the study drug and a known response pattern to it and cannot be otherwise explained by the patient's medical condition or concomitant medication
- probably related: meets all criteria mentioned above and has to improve after dechallenging the patient with the study drug.
- possibly related: an AE that has a temporal relationship between administration of the study drug and its occurrence and is a known response pattern to the IMP but could also be explained by the patient's medical history or treatment.
- Unrelated: an AE without a relationship in time to study drug treatment and which is most likely explained by the patient's medical condition or therapies.

## 8.10 Recording, Reporting, and Follow-Up Procedures

# 8.10.1 Procedures for Recording, Reporting, and Follow-Ups of Adverse Events

#### **Recording and Reporting of Adverse Events**

The patient will be given the opportunity to report AEs spontaneously at every on-site visit and telephone call. Moreover, the rater will propose an open-ended, non-leading question to the participant to detect AEs.

Documentation needs to be done in the patient's medical record and in a special section for adverse events in the CRF where the following details must be entered:

- Type of adverse event (diagnosis or syndrome; if not known signs or symptoms)
- Start (date)
- End (date)
- Severity (mild, moderate, severe, life-threatening/disabling, death)
- Serious (no / yes)
- Unexpected (no / yes)
- Outcome (resolved, ongoing, ongoing improved, ongoing worsening)
- Action taken (none, study medication dose reduced, study medication interrupted, study medication discontinued, medication therapy, surgical procedure, hospitalization, other)
- Relation to study drug (possibly, probably or definitely related or not related)

The investigator should use syndromes or diagnosis of standard medical terminology to record adverse events, whenever possible.

The Sponsor should be informed immediately by the investigator on-site, if an AE is thought to be at least probably related to the study drug treatment to discuss whether or not the administration of the IMP should be stopped.

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

Serious adverse events

#### Pregnancies

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e. no more than 24 hours after becoming aware of the information). New significant information includes the following:

- New signs or symptoms or a change in the diagnosis.
- Significant new diagnostic test results.
- Change in causality based on new information.
- Change in the event's outcome, including recovery.
- Additional narrative information on the clinical course of the event.

Investigators must also comply with local requirements for reporting SAEs to the local health authority and IRB/EC.

#### **Follow Up of Adverse Events**

An AE will be followed until the patient has recovered/ it has resolved, has reached a stable state, the investigator determines that it is no longer clinically significant, or the patient is lost to follow up. The end of an AE should be documented in the CRF and the patient's record. If an AE is still ongoing at the end of the study for a patient, follow up will be provided until resolution/stable level is achieved, or until it no longer is clinically significant by the judgement in the investigator, or until the patient is lost to follow up. In the latter the investigator has to take all possible actions in the discretion of his judgement to contact the patient and document a loss of follow-up in the source documents.

In case of withdrawal from the study due to an AE, an Early Termination (ET) Visit will be scheduled as soon as possible followed by a Safety Follow-Up Visit after 2 weeks + 2 days of the ET (if the ET is performed after 5 days after the last intake of study drug).

# 8.10.2 Recording, Reporting, and Follow-Up Procedures for Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions

# Reporting and Recording of Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions

Investigators will seek information on SAEs and SUSARs at each patient contact throughout the trial. As for all AEs, whether reported by the patient or noted by study personnel, SAEs and SUSARs will be recorded in the patient's medical record and on the Adverse Event Section of the CRF.

In the event of a **serious adverse event**, the investigator has to use all supportive measures for best patient treatment. An SAE form must be completed by the investigator and reported no more than 24 hours after receiving notice of the event.

The site must provide the Sponsor with a detailed description containing at least the symptoms and course of events, the actions taken, the medication given and if the dose of the study drug was changed. The following details should be available with the initial report:

- Patient number
- Patient: date of birth, ethnic origin
- Name of investigator and investigating site
- Period of administration
- The suspected investigational medicinal product (IMP)
- The adverse event assessed as serious
- Concomitant disease and medication
- Relevant medical history
- Short description of the event and outcome
- Description
  - o Onset and if applicable, end
  - Therapeutic intervention
  - Causal relationship to each of the study drugs (for definition see: 8.2.1.)
  - o Hospitalization or prolongation of hospitalization
  - o Death, life-threatening, persistent or significant disability or incapacity

This insight from the investigator is very important for the Sponsor to assess the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

In case of a new development of the event, the initial report should be followed by the followup report, indicating the outcome of the SAE.

A copy of the reports will be provided to AOP Orphan Pharmaceuticals for safety records.

**SUSARs** need to be reported and followed up in the same manner as SAEs. The Sponsor decides if the event needs to be classified as a SUSAR in discussion with the investigator. Therefore, detailed information about the event and the subsequent actions should be made available within 24 hours by the investigator and any relevant updates should be reported within 24 hours. SUSARs will be reported to the required regulatory authorities, investigators/institutions, and ethical committees in compliance with all reporting requirements according to local regulations and good clinical practice by the Sponsor and/or its designees.

After informed consent has been obtained but prior to initiation of the study drug, only SAEs considered to be related to a protocol-mandated intervention should be reported (e.g. SAEs related to invasive procedures such as withdrawal of blood).

#### Follow Up of Serious Adverse Events and SUSARs

For SAEs, SUSARs and pregnancies, the Sponsor or a designee may follow up by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details and outcome information (e.g. from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case. An SAE and SUSAR will be followed until it has resolved, has reached a stable state, the investigator determines that it is no longer clinically significant, or the patient is lost to follow up.

If an SAE or SUSAR of a participant is still ongoing at the end of the study, follow up will be provided until resolution/ a stable level is achieved, or until the SAE or SUSAR is no longer clinically significant by the judgement in the investigator, or until the patient is lost to follow up. In the latter the investigator has to take all possible actions in the discretion of his judgement to contact the patient. A loss of follow-up should be documented in the source documents.

In case the IMP was withdrawn due to an SAE or SUSAR, patients will be advised to come to the hospital as soon as possible for an Early Termination Visit (see 5.7). A Safety Follow-Up Visit should be performed 2 weeks + 2 days after the last intake of study medication (if the Early Termination Visit occurs not longer than 5 days after the discontinuation of the study medication). (see 5.6) The patient should be followed up until he/she has recovered/ it has resolved, has reached a stable state, the investigator determines that it is no longer clinically significant, or the patient is lost to follow up.

# 8.11 Review and Annual report on Adverse Events, Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions

Data from this study will be reviewed periodically by the Sponsor or a designee to detect any safety concern(s) related to the study drug as early as possible so that the investigators, regulatory authorities, and IRB/IEC will be informed appropriately and as early as possible. SAEs will be reviewed ongoing and reconciliations will be performed in collaboration with the Sponsor of the study.

If necessary, additional safety measurements can be implemented during the course of the

study after approval by the local IRB/IEC and regulatory authorities.

Once per year, the Sponsor or principal investigator will supply a report on the safety of trial subjects with all available relevant information concerning patient safety during the reference period to the competent supreme federal authority where the trial is being conducted. This report will also be supplied to the responsible ethics committee.

The annual safety report will be compiled according to the corresponding ICH guideline E2F "Development Safety Update Report – DSUR".

The data lock point for the patient data to be included and analyzed is the day of the overall approval of the clinical trial.

The Sponsor or principal investigator will supply the report within 60 days of one year after the reference date (data-lock point).

#### 9 Documentation

The accomplishments of the study in agreement with the GCP-guidelines and the investigational plan as well as the accuracy of all data documented in the CRF are the responsibility of the Investigator. All collected data of this study have to be recorded on the CRF and/or the patient's record by appropriate authorized persons. This also includes data of patients who dropped-out of the study. It has to be assured that all persons authorized for CRF entries can be identified. A list with signatures and identification codes of the persons must be archived in the ISF and TMF. Moreover, logs according to ICH E6 (e.g. Signature/Delegation/Screening/Drug Accountability log) will be implemented and maintained by the investigator.

The investigator records the participation of a patient on a special identification list of patients (Screening Log). This list gives the possibility for a later identification of the patients and contains the patient number, full name, date of birth and the date of the enrolment into the study. The identification list of patients remains in the study center after the closure of the study. Additionally, the participation of the patient in this clinical study has to be recorded in the patient's medical record.

Each patient will receive a unique patient identification number. Data will be documented using this code for each patient that will also be used for communication with the Sponsor and other authorities. Only the Investigator and his/her designees will be able to connect the number and the patient's name. Data collection must be completed for each subject which has signed an ICF and was administered study drug.

Patient's data will be stored on-site in a locker to which only the investigator and his/her designees have access. Personal patient information (such as name, date of birth etc.) is stored separately from the research data.

For all work involving data collections of human information, electronic or otherwise, the study centre will adhere to the law as laid down in the European Regulation (EU) 2016/679 (Regulation (EU) of the european parliament and of the council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation)) as well as national data protection law. Adequate measures to ensure data protection, confidentiality will be duly taken into account by the Investigators and all parties involved in the study.

# 9.1 Data Recording (Case Report Form, CRF and Patient's Record)

In this study, a Case Report Form (CRF) will be used for direct entry of the assessments of the scales used and for the telephone calls. Demographic data, medical history, neurological and PD history, medication history (including anti-parkinson's disease medication), adverse events (including SAEs, SUSARs, ADRs), concomitant medication, the assessments of Vital Signs, and the neurological and physical examination will be provided at the Screening / Baseline Visit in the CRF. The patient's record will be used to document the date and identification of the visit, the investigator(s) conducting the visit, the process of Informed Consent (the description of the process of informed consent, the person conducting Informed Consent, the date, time, and version of ICF), the time and date of all the assessment of the clinical scales, the time and date of urine pregnancy tests, protocol deviations (including actions), and the Drug Accountability (for returned and assigned kits).

The CRFs and the patient's records are established to implement the Clinical Study Protocol, to facilitate subject observation and to record subject and IMP data during the clinical investigation according to the trial's protocol. In this study, they exist as printed or written documents and are direct-entry CRFs.

In the patient's record and the CRFs, the following data should be documented:

- the date and identification of the investigation, including the version number of the Clinical Study Protocol;
- identification of the subject, date of enrolment, demographic data (at the Screening / Baseline Visit);
- identification of the IMP by lot number and kit number (if applicable);
- medical diagnosis for which the subject is to be treated with the IMP to be investigated together with any concomitant illness (at the Screening / Baseline Visit);
- subject compliance information for concurrent procedures measures and for any emergency;
- relevant previous medication and/or procedures (at the Screening / Baseline Visit only);
- (changes to the) subject baseline characteristics (at the Screening / Baseline Visit only):
- concomitant medication and/or procedures;
- compliance with the inclusion/exclusion criteria;
- dated clinical and non-clinical findings according to the Clinical Study Protocol;

- procedural data;
- subject assessment during the use of the IMP and follow-up with dates;
- reported adverse events and adverse effects with dates;
- date of the end of follow-up;
- signature(s) of the clinical investigator(s) at the completion of follow-up

Therefore, the CRF and the medical record of the patient will be a source document in this study.

Only the use of ballpens is allowed for the entry in paper-based records. Corrections have to be made in a way, that the previous entries remain readable (the use of any instrument of correction is not allowed). Corrections have to be signed and dated by the authorised person, who made the corrections. Data, which are not available or were not collected, have to be clearly identifiable as such (NA). The reasons should be documented, if necessary. The investigator assures, that all data of patients are recorded immediately, readable, completed, and correct in the patient's chart and in the CRFs.

After the end of the study (end of the study defined as the last visit of the last patient) and after the verification regarding the plausibility and completeness by the Monitor, all documents and data relating to the study will be kept in an orderly manner by the investigator in a secure study file. Source data will be stored for 30 years (for medical records and other original data) after the end of the study (i.e. last visit of the last patient) according to local and national regulatories. It is the responsibility of the investigator to inform the Sponsor before study related documents will be destroyed.

Monitors, auditors, and other authorized agents of the Sponsor or its designee, the EC/IRB approving the research, local law regulatory agents and appropriate authorities in conducting investigations for which the person's medical history is necessary will be granted access to the study subject's original medical records without violating the confidentiality of the subject to the extent permitted by the law and regulations. In any presentation of the results of this study or in publications, the subject's identity will remain confidential.

#### 9.2 Trial Folders

The trial folders should serve as gapless documentation. Individually or together they should allow the evaluation of the trial implementation as well as quality of data.

#### 9.2.1 Trial Master File (TMF)

The paper-based TMF, established at the beginning of the trial and secured in a safe place, contains all essential documents that demonstrate that the trial is conducted in accordance

with regulatory requirements and ICH GCP. All documents will be maintained and updated as appropriate throughout the trial. Previous versions of the documents must be retained in the TMF and will be clearly labelled as outdated. Previous versions will be relocated in a section for outdated documents. The TMF is archived at the end of the study for 15 years.

#### 9.2.2 Investigator Site File (ISF)

The paper-based ISF, established at the beginning of the trial will be secured in a safe place (the file is provided to the site at the site initiation visit). It contains all essential documents maintained by the PI. All documents will be maintained and updated as appropriate throughout the trial. Previous versions of the documents must be retained in the ISF and will be clearly labelled as superseded-previous versions will be relocated in a section for outdated documents. Within each monitoring visit, the ISF will be checked for actuality and completeness in accordance to the formalities. After completion or discontinuation of the study this ISF has to be kept for 15 years.

## 9.3 Data Storage

#### 9.3.1 Storage duties of the Sponsor

The Sponsor has to keep all study-relevant documents of the clinical study after completion or discontinuation of the study for a minimum of 15 years.

## 9.3.2 Storage duties of the investigator

The Investigators have to keep all records and documents, which are related with the study or the allocation of investigational medicinal products (e.g. data entry form, consent form, list of the allocations of investigational medicinal products and further relevant documents), for a minimum of 15 years. Medical records and other source data (e.g. paper-based CRF) have to be kept for 30 years.

# 10 Data Management

Data are administered and processed by members of the study team with the support of the software Microsoft Word, Excel, and IBM SPSS Statistics.

The evaluation of the data takes place by the programmed range-, validity- and consistence checks. In addition to that a manual/visual evaluation of the plausibility in accordance with the requirements of the GCP is performed. Queries may occur, which will be forwarded to the investigator by the Monitor of the study. By means of the queries the investigator has to evaluate and respond to the accrued discrepancies. After the record of all entries and clarification of all queries, the data based will be closed at the completion of the study. This performance has to be documented.

#### 11 Protocol Deviations

All deviations to the study protocol have to be documented in the patient's record with the explanation for variance. Deviations have to be announced to the Sponsor, who is responsible for their evaluation, within 24 hours after receipt of knowledge. The report should include the patient's study code, sex, year of birth, a brief description of the event, the cause of it (if applicable), the time, the date, the duration of the event, and the corrective and preventive measurements performed. Protocol Deviations will be reported to the Sponsor to decide if the patient will be discontinued in the study or not.

The Sponsor can terminate a trial during the course of it, whenever a reason for concern appears. The Sponsor or the investigator can discontinue a patient's participation in the trial on their behalf (for criteria see 4.3). Reasons for termination of a trial or of a study participant have to be documented in the patient's record or other source documents. In case of a security termination, the test person has to be further monitored. Deviations have to be analyzed whether changes of the clinical investigation plan or the closure of the study are necessary. If necessary, the ethics committee or the responsible authorities have to be informed.

In case of a withdrawal from the study, the data will be included in the analysis up to the time of discontinuation.

# 12 Statistical Analysis

## 12.1 Determination of Sample Size

This is an open-label study. The sample size for this study is not based on statistical considerations; Up to 48 subjects who completed the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and met patient exclusion/inclusion criteria will be enrolled.

In the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study a total of 38 patients (19patients per group) provided 80% power at two-sided 5% significance level to detect a statistically significant difference in the change from baseline to Termination visit in MDS-UPDRS Part I score between nabilone and placebo assuming a true difference of 2.5 points. This sample size calculation assumed a standard deviation of the change from randomization to week 4 to be 2.4 points. (46) With a drop- out quote of 25 % we planned to include 48 patients in the trial. We chose this design because it has the advantage that the patient population enrolled is enriched by including only responders. (48) The sample size calculation for the NMS-Nab Study was performed with the Program nQuery Advisor (Version 7).

# 12.2 Study Populations: Datasets or Populations analyzed

Safety and tolerability summaries will be based on a safety set which will include all patients receiving at least one dose of study medication and completing at least V 1 will be analysed. The safety set will be used for summaries of safety and tolerability. Additionally, summaries of baseline and demographic data will be produced out of the safety set. The efficacy analysis for the secondary endpoints will also be performed including all screened subjects with at least one Visit after the V 0. All summaries for efficacy will be based on the set.

In case of a drop-out, no interpolation can be performed. Therefore, the primary analysis is a per-protocol analysis.

## 12.3 Background and Demographic Characteristics

All baseline and demographic summaries will be produced for the data of patients gained at the Screening / Baseline Visit out of the safety dataset.

The number and characteristics of patients in the safety set, , the number of AEs, SAEs and SUSARs with description, the number of subjects with premature discontinuation from the study/or the study drug along with reasons for discontinuation will be provided. Furthermore, the number of screened subjects, the number of screening failures and reasons why they have been excluded will be given.

A consort diagram will be provided.

## 12.4 Safety Analysis

This is a phase III open-label trial to evaluate the long-term safety and tolerability of nabilone for non-motor symptoms of patients with PD. Data analysis will be performed using IBM SPSS Statistics Software and Microsoft Excel.

The primary safety analysis will be performed with the safety data set. Additionally, a safety analysis will be performed on all events as well as the hallucination item, orthostatic hypotension item and day-time sleepiness item of Part I of MDS-UPDRS occurring through the overall study. This will be a descriptive analysis reporting overall number and frequencies of the item's points score, AEs, SAEs, and SUSARs in patients taking nabilone.

Separate summaries of AEs in regard of severity and relationship to the study drug, separate summaries of AEs leading to withdrawal from the study and separate summaries for SAEs will be provided.

Tolerability measures will be provided in a descriptive analysis and will include the number of patients who discontinued from the study (%) and the number of patients who discontinued from the study due to an AE (%).

Safety measures include vital signs including performance of active orthostatism, the hallucination item (1.2, 0-4 points) of MDS-UPDRS Part I, the orthostatic hypotension item (1.12, 0-4 points) of MDS-UPDRS Part I, the Daytime sleepiness item (1.8, 0-4 points) of MDS-UPDRS Part I, and the C-SSRS. All patients will therefore be questioned about the occurrence of an AE at each scheduled and unscheduled on-site visit or telephone visit. Vitals signs including performance of active orthostatism will be taken at any scheduled visit on-site. (see 7.2) In the latter the heart rate and blood pressure of the patient will be measured after 10 minutes of quiet resting in a supine position and at 1, 2, 3, 5, and 10 minutes - time points of active standing.

Clinical examination and aurine pregnancy test for women of childbearing potential will be executed at the Screening / Baseline Visit, the Visits V 1, V 2, V 3, an Early Termination Visit (if applicable), and the Safety Follow-Up Visit (except for urine pregnancy test).

## 12.5 Efficacy Variables and Analysis

Results of the changes of all clinical scales in this trial will be shown in a descriptive way by median and interquartile range (quartile 1, quartile 3) f. Mean and standard deviation for the descriptive analysis will also be provided. P-values for the change of the results will be given. The secondary efficacy criteria will be measured as the change in all clinical scales and questionnaires between V 1 and month 6, except for the MMSE and the MoCA. The changes of these scales will be measured as the change between the Screening Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study and the month 6 visit (V 3) of this study. For the study's secondary efficacy analyses, mean changes from V 1 (or the Screening Visit of the NMS-Nab study for MMSE and MoCA) to the 6 months visit will be analyzed by Wilcoxon matched-pairs test. (49) For all analyses, statistical significance will be set at the 2-sided 5% level. To estimate the treatment effect, we will then compare mean change from V 1 to month 6 visit using analysis of covariance, with value at V 1 as covariate and the treatment group as main effect.

Because an interpolation of data will not be performed in case of a drop-out, the primary analysis is a per-protocol analysis.

Moreover, sensitivity to treatment will be assessed using effect sizes of the different outcome variables when using nabilone to treat non-motor symptoms in Parkinson's disease.

For CGI-I analyses, distributions of aggregated ratings (amelioration, aggravation) after 6 months will be analyzed with the Wilcoxon matched-pairs test. (49)

# 12.6 Exploratory Endpoint

For the Eye-tracking analyses, mean changes from the evaluations of the Screening and the Termination Visit of the randomized placebo-controlled, double-blind, parallel-group, enriched enrolment randomized withdrawal study to V 2 of this study will be compared using the Wilcoxon matched-pairs test.

# 12.7 Handling of Missing Data

After early withdrawal of study drug treatment, all patients will perform an ET visit. All withdrawals from the study or the study drug will be included in the safety analysis up to the

| time of discontinuation regardless of the duration of their participation. In case of a drop-out, no interpolation can be performed. Therefore, the primary analysis is a per-protocol analysis. |
|---|

# 13 Quality Management

Training, monitoring and audits are performed for quality assurance reasons within this clinical study. Monitoring and auditing procedures developed or endorsed by the Sponsor will comply with ICH-GCP guidelines and local legal requirements to ensure acceptability of the study data and patient's safety.

#### 13.1 Qualifications

The Sponsor is responsible for selecting the investigator and Institution. Each investigator should be qualified by training and experience and should have adequate resources. Each individual involved in conducting a trial should be qualified by education, training and experience to perform his or her respective task(s) (see ICH GCP E6).

To meet those objectives, every member of the study team must be GCP-trained. A Certificate of MDS-UPDRS Training, a C-SSRS Training Certificate, and experience in using the other scales (e.g. MMSE) must be provided by every investigator in the trial who intends to use these scales. The members of the study team must be trained on the trial's protocol and the completion of the source data entry (CRF and patient's record) by the principal investigator or an authorized designee. This process has to be documented in the ISF. Authorization of a member of the study team to perform study related tasks have to be reported in the Delegation Log of the ISF.

# 13.2 Monitoring

A study monitor will perform source document verification at regular intervals in accordance with GCP and ICH guidelines. The objectives of the monitoring procedures are to ensure that the trial subject's safety and rights as a study participant are respected, that accurate, valid and complete data are collected, used, and stored, and that the trial is conducted in accordance to the trial protocol, the principles of GCP and local legislation.

All investigators agree that the monitor regularly visits the trial site. For monitoring, all study-related documents must be given access to the monitor by the investigator for confirmation of data. Moreover, the investigators assure that the Monitor will receive appropriate support in their activities at the trial site, as agreed in separate contracts.

The Informed Consent Form (ICF) includes a statement that the Monitor has the right – while observing the provisions of data protection legislation – to compare CRFs with the trial subject's medical records (doctor's notes etc.).

A study specific monitoring plan will be established and the study will be monitored with the agreed plan.

All representatives from regulatory authorities and the EC/IRB will be gained access to the study-related documents needed for their investigation. Protection of the patient's personal data will be guaranteed to the extent possible.

## 13.3 Audits and Inspections

During the course of a study, a Quality Assurance audit or inspection can be performed by regulatory authorities, the ethics committees, or the Sponsor's delegates. Therefore, the investigator has to grant direct access to all data and must provide support at all times. The aim of an audit is to verify the validity, accuracy and completeness of data, to establish the credibility of the clinical trial, and to check whether the trial subject's rights and trial subject safety are being maintained. The Sponsor may assign these activities to persons otherwise not involved in the trial (Auditors). These persons are allowed access to all trial documentation (especially the trial protocol, CRFs, trial subject's medical records, drug accountability documentation, and trial-related correspondence).

After each external audit an audit-certificate by the Auditor has to be delivered to the investigator. This certificate has to be kept in the ISF to evidence the audit to the regulatory authorities in the case of an inspection by them. The audit-report is delivered to the Sponsor of the study. An audit-certificate will be attached to the final report at the end of the study. Additionally, according to the Austrian Medicines Law (AMG) audits and inspections by regulatory authorities may be performed.

All persons conducting audits undertake to keep all trial subject data and other trial data confidential.

# 14 Reporting

## 14.1 Annual Progress Reports

The Sponsor/investigator will submit a summary of the progress of the trial to the accredited EC and to the competent supreme federal authority (if applicable) once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, data of safety of the trial subjects including serious adverse events/ serious adverse reactions, other problems, protocol deviations and amendments.

The annual safety report will be compiled according to the corresponding ICH guideline E2F "Development Safety Update Report – DSUR".

The data lock point for the patient data to be included and analyzed is the day of the overall approval of the clinical trial. The Sponsor or principal investigator will supply the report within 60 days of one year after the reference date (data-lock point).

## 14.2 Final Study Report

The end of the study is defined as the last visit of the last patient of the study (LPLV). On completion of the study, the EC/IRB, and the regulatory authorities will be notified that the study has ended. Within one year after the end of the study, the investigator/Sponsor will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited EC/IRB.

All information regarding this clinical study has to be kept in confidence. The statistical analysis and the integrated final study report will be prepared according to ICH E6 and finalized within 12 months after the last patient's last visit (LPLV) took place. The final study report will be reviewed and signed by the Sponsor, the principal investigator and all further responsible persons. All information in that report is strictly confidential.

The principal investigator will sign the final study report of the clinical trial. This confirms that the report describes implementation and results of the clinical trial by the best of his knowledge.

#### 15 Publication

The results of this study will be published according to the principles of publication policy. There are no arrangements on publication issues with subsiding parties.

#### 16 Amendments

Amendments must be submitted to the appropriate regulatory authorities and ethical committees. Substantial amendments may be implemented only after approval of both parties has been obtained. Urgent amendments that are intended to eliminate an apparent immediate hazard to subjects may be implemented prior to receiving approval. However, approval must be obtained as soon as possible after implementation. Therefore, the Sponsor or its designee must inform the regulatory authority and the EC about the new events, the measures taken and their plan for further action as soon as possible. The procedure should be held as follows: immediate telephone contact, followed by an e-mail or FAX notice, followed by a follow-up letter.

# 17 Ethical and Regulatory Aspects

#### **Ethical Conduct of the Study**

Ethics committee (EC) authorization for this study will be required. The project raises important issues of consent, confidentiality, data security, quality control, and national data protection legislation. To protect the information on each participating individual, protect privacy, and prevent misuse of data, all investigators and all parties involved in this study will adhere to national codes and rules for working with participant's clinical data. Participants will be labeled in a coded fashion with unique identifiers. Data will be held secure and confidential and kept apart from personal identifiers.

The project will be conducted in strict adherence to the Convention for the Protection of Human Rights and Fundamental Freedoms, and EU regulations on ethical issues including the Regulation (EU) 2016/679, and the Directives 2001/20/EC, and 2005/28/EC relating to implementation of good clinical practice in the conduct of clinical trials.

#### **Regulatory Requirements**

The present study will be conducted in compliance with Good Clinical Practices (ICH-E6: GCP recommended for adaptation on 1st of May 1996 by the ICH Steering Committee), the Declaration of Helsinki in its latest version concerning the conduct, evaluation and documentation of the study, the "Charter of Fundamental Rights" of the European Union (2000/C 364/01), the local laws and regulations and the applicable regulatory requirements.

When conducting a clinical trial on drugs for use in humans in Austria the Medicines Act ("Arzneimittelgesetz", AMG) has to be considered. This Act implemented the European Directives 2001/20/EC and 2005/28/EC into national law. In particular, section III (Clinical Trials) is relevant for the conduction of a clinical trial.

## 17.1 Responsibilities of the Sponsor and the investigator

The Sponsor of this clinical trial will assume responsibility for inducement and organization of the implementing trial according to the AMG. The procedures set out in this study protocol are designed to ensure that the Sponsor and the investigator abide the principles of ICH E6 recommended for adaptation on 1st of May 1996 by the ICH Steering Committee and the Declaration of Helsinki concerning the conduct, evaluation and documentation of the study. The study will also be performed adhering the local legal conditions and requirements. Each investigator has to confirm this by signing the study protocol.

Responsibilities of the Sponsor:

- Verification of the understanding of the Investigator's Brochure or the described study medication
- Verification of the understanding of treatment schedule
- Ensuring for enough time and capacity for the implementation of this study
- Correct collection and documentation of data, reporting
- Provision of all data to the Sponsor, monitor or relevant authorities for audits or inspections
- Assurance for the confidential handling of patient's data and information

The principal investigator accepts the responsibility for the implementation of this clinical trial at this study site according to the AMG.

## 17.2 Approval and Consent

#### **Independent Ethics Committee or Institutional Review Board**

Before initiation of the study, the conduct of the study will be submitted to our local Ethics Committee (EC) / Institutional Review Board (IRB). Written approval of the study, the protocol, the Informed Consent Form (ICF), all questionnaires, and all other relevant study documentation must be obtained before the first patient will be screened and the study drug is released to the investigator. Any necessary extensions or renewals of EC/IRB approval must be obtained for changes to the study such as amendments to the protocol, the ICF or other study documentation. The written approval of the EC/IRB together with the approved ICF must be filed in the study files.

The investigator will report promptly to the EC/IRB any new information that may adversly affect the safety of the participants or the conduct of the study. The investigator will submit written summaries of the study status to the EC/IRB as required. On completion of the study, the EC/IRB will be notified that the study has ended. End of the study is the time when the last visit of the last patient has been performed (LPLV).

#### **Regulatory Authorities**

All relevant study documentation will be submitted to the regulatory authorities according to local/national requirements, for review and approval before initiating the study.

On behalf of the AMG in Austria, the Sponsor of the clinical trial submits the application to the competent ethics committee (EC) and the competent authority (CA). The CA reviews only the justification for and the relevance of the Clinical Trial. The EC acts as the "expert reviewer" for the CA and decides within 35 days, with only one "clockstop" possible to obtain supplementary information. If the EC vote is negative, the CA issues a legal document ("Bescheid") prohibiting the clinical trial.

On completion of the study (LPLV), the regulatory authorities will be notified of the end of the study.

#### **Informed Consent**

The process of obtaining informed consent must be in accordance with applicable regulatory requirement(s) and must adhere to GCP.

No subject will undergo any study related examination or activity in the responsibility of the investigator before he/she has given written informed consent to participate in the study. The investigator or designee explains orally and in writing manner the nature, the duration, the importance, the relevance, the purpose of the study, the consequences, and the action of the drug in such a manner that the patient and a study partner (if applicable) are aware of potential risks, inconveniences, and adverse events of the study and the study drug. It should also be straightened out that the subject is free to choose to take part in the study or to withdraw from participation without consequences for his/her further care. The patient should be given the opportunity to ask for clarification of any points he/she does not understand and, if necessary, ask for more information. At the end of the interview, the subject will be given ample time to consider his/her participation in the study. Subjects and the investigator will be required to sign and date the ICF. After signatures are obtained, the ICF will be kept and archived by the investigator in the investigator's site file. A signed and dated copy of the Patient Information and Informed Consent Form will be provided to the patient. If new information becomes available that may be relevant to the subject's willingness to continue participation in the study, a new ICF will be approved by the EC/IRB (and regulatory authorities, if required). The study subjects will be informed about this new information and re-consent will be obtained.

#### **Risks and Benefits**

**Benefits:** The patients participating in the study will receive specialized care and regular clinical monitoring. The results of this trial will be useful to evaluate the long-term safety, tolerability and effects of nabilone on non-motor symptoms in PD. Moreover, management of NMS are an important area of unmet need in PD. Due to the overall impact of NMS in PD and based on the influence of the endocannabinoid system on NMS in broad manner in PD, we perform this trial of nabilone in PD patients. Hopefully, a symptomatic improvement of the patient's clinical condition could be achieved.

**Risks:** Disadvantages of participation could be the additional time spent in the hospital, currently unknown risks of the study drug therapy, or allergies to components of the IMP the patient is unaware at inclusion in the study.

Treatment care in the study population will not be affected by the trial because nabilone will be used as an add-on therapy.

Generally, nabilone is well tolerated. In this trial we will only include patients that participated in the NMS-Nab Study and had no drug-related SAE or moderate or severe AE. Therefore, the risk of allergic reactions to components and SAEs related to the drug are minimized. Common adverse reactions (>1/100 to <1/10) observed in patients are somnolence, vertigo, euphoria, ataxia, impaired vision, difficulties to concentrate, sleep disturbances, dysphoria, a headache, hypotonia, nausea, and a dry mouth. Controlled trials with patients taking nabilone showed that at least one side effect occurred per subject. Most patients develop a tolerance in regard of adverse events concerning the CNS and therefore somnolence and euphoria reside after some weeks. This effect is reversible. The potential to cause mental addiction is unknown and no patient has shown withdrawal symptoms in clinical trials. Minor risks of nabilone (>1/10.000 to <1/1.000) include confusion, disorientation, hallucination, psychosis, depression, difficulties in coordination, tremor, loss of appetite, anxiety, depersonalisation, tachycardia, and abdominal pain.

All AEs will be rapidly detected by close clinical monitoring. In case of an AE the patient should be followed up until he/she has recovered/ it has resolved, has reached a stable state, the investigator determines that it is no longer clinically significant, or the patient is lost to follow up. Study treatment will be stopped in the discretion of the investigator and appropriate measurements, reporting, and visits on-site will be performed.

These controlled risks must be balanced against the prospect of identifying a new therapeutic option for non-motor symptoms in PD. All patients are not naïve to the investigational treatment.

There are no known risks in relation to the Eye-tracking analysis.

#### 17.3 Patient Insurance

During their participation in the clinical trial the patients will be insured as defined by legal requirements. The Sponsor is providing insurance in order to indemnify (legal and financial coverage) the investigator/trial center against claims arising from the study, except for claims that arise from malpractice and/or negligence. The compensation of the subject in the event of study-related injuries will comply with the applicable regulations.

This insurance covers for damage to research subjects through injury or death caused by the study. The insurance applies to the damage that becomes apparent during the study.

## 17.4 Data Protection and Confidentiality

All local legal requirements regarding data protection will be adhered to. All study findings and documents will be regarded as confidential. The investigator and members of the

research team must not disclose any information without prior written approval from the Sponsor. The pseudonymity of patients participating must be maintained. Throughout documentation and evaluation, the patients will be identified on CRFs and other documents by an ascending number according to their order of screening. Documents that identify the patient personally (e.g., the signed informed consent, patient identification list, patient's record) must be maintained in confidence by the investigator. The patients will be informed in the ICF that all study findings will be stored in a locked cabinet and on computer and handled in strictest confidence.

## 17.5 Discontinuation of the Study by the Sponsor

The Sponsor or its representative is authorized to temporary hold or discontinue the study for any reason and at any time decided.

The investigator/Sponsor will notify the accredited EC/IRB of the end of the study (LPLV). The Sponsor or its representative will notify the EC/IRB immediately of a temporary halt of the study, including the reason of such an action. In case the study is ended prematurely, the Sponsor or its designee will notify the accredited EC/IRB within 15 days, including the reasons for the premature termination.

#### 18 References

- 1. Iannotti FA, Di Marzo V, Petrosino S, *Endocannabinoids and endocannabinoid-related mediators: Targets, metabolism and role in neurological disorders.* Progress in lipid research, 2016. 62: p. 107-128
- 2. Hui-Chen, Mackie K, *An Introduction to the Endogenous Cannabinoid System*. Biological Psychiatry, 2016. 79: p. 516-525
- 3. Turu G, Hunyady L, Signal transduction of the CB1 cannabinoid receptor. J. Mo Endocrinol, 2010. 44: p. 75-85
- 4. Di Marzo V, De Petrocellis L, *Why do cannabinoid receptors have more than one endogenous ligand?.* Philos Trans R Soc Lond Ser B Biol Sci, 2012. 367: p. 3216-3228
- 5. Stella N, Cannabinoid and cannabinoid-like receptors in microglia, astrocytes, and astrocytomas. Glia, 2010. 58: p. 1017-1030
- 6. Matias I, Di Marzo V, *Endocannabinoids and the control of energy balance*. Trends Endocrinol Metab, 2007. 18: p.27-37
- 7. Izzo AA, Cannabinoids and intestinal motility: welcome to CB2 receptors. Br J Pharmacol, 2004. 142: p. 1201-1202
- 8. Pertwee RG, Receptors and channel targeted by synthetic cannabinoid receptor agonists. Curr Med Chem, 2010. 17: p. 1360-1381
- 9. Melis M, Pistis M, Endocannabinoid signaling in midbrain dopamine neurons: more than physiology?. Curr. Neuropharmacol., 2007. 5: p. 268–277
- 10. Maccarrone M, Gubellini P, Bari M, Picconi B, Battista N, Centonze D, et al., Levodopa treatment reverses endocannabinoid system abnormalities in experimental parkinsonism, J. Neurochem, 2003. 85: p. 1018–1025
- 11. García C, Palomo-Garo C, García-Arencibia M, Ramos J, Pertwee R, Fernández-Ruiz J, *Symptom-relieving and neuroprotective effects of the phytocannabinoid Δ-THCV in animal models of Parkinson's disease*. Br J Pharmacol, 2011. 163: p. 1495–1506
- 12. Kluger B, Triolo P, Jones W, Jankovic J, *The Therapeutic Potential of Cannabinoids for Movement Disorders*. Movement Disorders, 2015. 30, p. 313-327
- 13. Kalia LV, Lang AE, *Parkinson's disease*. The Lancet Neurology, 2015. 386(9996): p.896-912
- 14. Braak H, de Vos RA, Bohl J, Del Tredici K, Gastric alpha-synuclein immunoreactive inclusions in Meissner's and Auerbach's plexuses in cases staged for Parkinson's disease-related brain pathology. Neurosci Lett., 2006. 396: p.67-72. Epub Dec 2005
- 15. Braak H, Del Tredici K, Rüb U, de Vos RA, Jansen Steur EN, Braak E, Staging of

- brain pathology related to sporadic Parkinson's disease. Neurobiol Aging, 2003. 24: p.197-211
- 16. Poewe W, The natural history of Parkinson's disease. J Neurol., 2006. 253 Suppl 7: VII2-6
- 17. Hely MA, Morris JG, Reid WG, Trafficante R, Sydney Multicenter Study of Parkinson's disease: non-L-dopa-responsive problems dominate at 15 years. Mov Disord., 2005. 20: p.190-199
- 18. Hely MA, Reid WG, Adena MA, Halliday GM, Morris JG, The Sydney multicenter study of Parkinson's disease: the inevitability of dementia at 20 years. Mov Disord., 2008. 23: p.837-44. doi: 10.1002/mds.21956
- 19. Pfeiffer RF, *Non-motor symptoms in Parkinson's disease*. Parkinsonism Relat Disord., 2016. Suppl 1:S119-22. doi: 10.1016/j.parkreldis.2015.09.004. Epub 2015 Sep 3
- 20. Abbott RD, Petrovitch H, White LR, Masaki KH, Tanner CM, Curb JD, Grandinetti A, Blanchette PL, Popper JS, Ross GW, *Frequency of bowel movements and the future risk of Parkinson's disease*. Neurology, 2001, 57: p.456-462
- 21. Savica R, Carlin JM, Grossardt BR, Bower JH, Ahlskog JE, Maraganore DM, Bharucha AE, Rocca WA, *Medical records documentation of constipation preceding Parkinson disease: A case-control study.* Neurology, 2009, 73: p.1752-8. doi: 10.1212/WNL.0b013e3181c34af5
- 22. Mahlknecht P, Iranzo A, Högl B, Frauscher B, Müller C, Santamaría J, Tolosa E, Serradell M, Mitterling T, Gschliesser V, Goebel G, Brugger F, Scherfler C, Poewe W, Seppi K; Sleep Innsbruck Barcelona Group, *Olfactory dysfunction predicts early transition to a Lewy body disease in idiopathic RBD.* Neurology, 2015. 84: p.654-8. doi: 10.1212/WNL.0000000000001265. Epub 2015 Jan 21
- 23. Ross GW, Petrovitch H, Abbott RD, Tanner CM, Popper J, Masaki K, Launer L, White LR, Association of olfactory dysfunction with risk for future Parkinson's disease. Ann Neurol., 2008. 63: p.167-17
- 24. Aarsland D, Marsh L, Schrag A, *Neuropsychiatric symptoms in Parkinson's disease.*Mov Disorders, 2009. 24: p.2175-86. doi: 10.1002/mds.22589
- 25. Noyce AJ, Bestwick JP, Silveira-Moriyama L, Hawkes CH, Giovannoni G, Lees AJ, Schrag A. *Meta-analysis of early nonmotor features and risk factors for Parkinson disease*. Ann Neurol, 2012. 72:893-901. doi: 10.1002/ana.23687. Epub 2012 Oct 15
- 26. Iranzo A, Tolosa E, Gelpi E, Molinuevo JL, Valldeoriola F, Serradell M, Sanchez-Valle R, Vilaseca I, Lomeña F, Vilas D, Lladó A, Gaig C, Santamaria J, Neurodegenerative disease status and post-mortem pathology in idiopathic rapid-eye-movement sleep behaviour disorder: an observational cohort study. The Lancet Neurol, 2013. 12: p.443-53. doi: 10.1016/S1474-4422(13)70056-5. Epub 2013 Apr 3

- 27. Seppi K, Weintraub D, Coelho M, Perez-Lloret S, Fox SH, Katzenschlager R, Hametner EM, Poewe W, Rascol O, Goetz CG, Sampaio C, *The Movement Disorder Society Evidence-Based Medicine Review Update: Treatments for the non-motor symptoms of Parkinson's disease.* Mov Disorder, 2011. 26 Suppl 3:S42-80. doi: 10.1002/mds.23884.
- 28. Schrag A, Sauerbier A, Chaudhuri KR, *New clinical trials for nonmotor manifestations of Parkinson's disease.* Mov Disorders, 2015. 30: p.1490-1504. doi: 10.1002/mds.26415.
- 29. Chaudhuri R K, Schapira A HV, Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. The Lancet Neurology, 2009. 8: p. 464-474
- 30. Chaudhuri R K, Healy D G, Schapira A HV, *Non-motor symptoms of Parkinson's disease: diagnosis and management.* The Lancet Neurology, 2006. 5: p. 235-245
- 31. Di Marzo V, Melck D, Bisogno T, De Petrocellis L, *Endocannabinoids: endogenous cannabinoid receptor ligands with neuromodulatory action*. Trends Neurosci, 1998. 21: p. 521-528
- 32. Castillo PE, Younts TJ, Chavez AE, Hashimotodani Y, *Endocannabinoid signaling* and synaptic function. Neuron, 2012. 76: p.70.81
- 33. Marinez-Orgado J, Fernandez-Lopez D, Lizasoain I, Romero J, *The seek of neuroprotection: introducing cannabinoids*. Recent Pat CNS Drug Discov, 2007. 2: p. 131-139
- 34. Sagredo O, Garcia-Arencibia M, de Lago E, Finetti S, Decio A, Fernandez-Ruiz J, *Cannabinoids and neuroprotection in basal ganglia disorders*. Mol Neurobiol, 2007. 36: p. 82-91
- 35. Barrero FJ, Ampuero I, Morales B, et al., *Depression in Parkinson's disease is related to a genetic polymorphism of the cannabinoid receptor gene (CNR1)*. Pharmacogenomics J, 2005. 5: p.135-141
- 36. Zuardi AW, Crippa JA, Hallak JE, et al., *Cannabidiol for the treatment of psychosis in Parkinson's disease*. J Psychopharmacol, 2009. 23: p. 979–983
- 37. Venderova K, Ruzicka E, Vorisek V, Visnovsky P., *Survey on cannabis use in Parkinson's disease: subjective improvement of motor symptoms*. Mov Disord, 2004. 19: p.1102–1106
- 38. Lotan I, Treves TA, Roditi Y, Djaldetti R., Cannabis (medical marijuana) treatment for motor and non-motor symptoms of Parkinson disease: an open-label observational study. Clin Neuropharmacol, 2014. 37: p.41–44.
- 39. Chagas MH, Eckeli AL, Zuardi AW, Pena-Pereira MA, Sobreira-Neto MA, Sobreira ET, Camilo MR, Bergamaschi MM, Schenck CH, Hallak JE, Tumas V, Crippa JA, Cannabidiol can improve complex sleep-related behaviours associated with rapid eye

- movement sleep behaviour disorder in Parkinson's disease patients: a case series. Journal of Clinical Pharmacy and Therapeutics, 2014. 39: p.564–566
- 40. Carroll CB, Bain PG, Teare L, et al., Cannabis for dyskinesia in Parkinson disease: a randomized double-blind crossover study. Neurology, 2004. 63: p.1245–1250
- 41. Mesnage V, Houeto JL, Bonnet AM, et al. Neurokinin B, neurotensin, and cannabinoid receptor antagonists and Parkinson disease. Clin Neuropharmacol, 2004. 27: p.108–110
- 42. Sieradzan KA, Fox SH, Hill M, Dick JP, Crossman AR, Brotchie JM, *Cannabinoids* reduce levodopa-induced dyskinesia in Parkinson's disease: a pilot study. Neurology, 2001. 57: p. 2108–2111
- 43. Chagas MH, Zuardi AW, Tumas V, Pena-Pereira MA, Sobreira ET, Bergamaschi MM, Dos Santos AC, Teixeira AL, Hallak JE, Crippa JA, *Effects of cannabidiol in the treatment of patients with Parkinson's disease: An exploratory double-blind trial.*Journal of Psychopharmacology, 2014. 28: p.1088–1098
- 44. Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease, The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord., 2003. 18: p.738-750
- 45. Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group, *King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation*. Movement Disorders, 2015. 30: p.1623-1631, Epub 2015 Jun 11.
- 46. Poewe W, Hauser RA, Lang A, for the ADAGIO Investigators, *Effects of Rasagiline* on the Progression of Nonmotor Scores of the MDS-UPDRS. Movement Disorders, 2015. 30: p.589-593
- 47. ICH Expert Working Group, *ICH Harmonised Tripartite Guideline, Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A*. European Medicines Agency. Step 5 Version, dated June 1995
- 48. US Dept of Health and Human Services Food and Drug Administration. Guidance for industry: enrichment strategies for clinical trials to support approval of human drugs and biological products. Dec. 2012, http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM332181.pdf. Accessed October 09, 2016.
- 49. Biaggioni I, Freeman R, Mathias CJ, Low P, Hewitt LA, Kaufmann H, on behalf of Droxidopa 302 Investigators, *Randomized Withdrawal Study of Patients With Symptomatic Neurogenic Orthostatic Hypotension Responsive to Droxidopa.*Hypertension, 2015. 65: p.101–107, Published online 2014 Dec 10,

# 19 Index of Figures

| Figure 1: Schematic Diagram for participants | |
|-----------------------------------------------------------------|----|
| 20 Index of Tables | |
| Table 1: Drug classes for non-motor symptoms in PD | 34 |
| Table 2: Nabilone for non-motor symptoms in Parkinson's Disease | 44 |